#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for Study 205883: A multi-centre, one-arm prospective study to evaluate efficacy and safety of switching from Entecavir (ETV) to Tenofovir Disoproxil Fumarate (TDF) in Japanese chronic hepatitis B HBeAg-positive and HBV-DNA undetectable subjects |
| <b>Compound Number</b> | : | GSK548470 |
| <b>Effective Date</b> | : | 18-SEP-2018 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 205883.
- This RAP is intended to describe the Safety and Efficacy analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

## **RAP Author(s):**

| Approver | Date | Approval Method |
|---|---|---|
| PPD | | |
| Study Statistician/ Biostatistics Group 1,<br>Biomedical Data Sciences Department, Japan. | | |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# RAP Team Approvals: Approved by (Approvals captured electronically in CARS system):

| Approver | Date | Approval<br>Method |
|---|---|---|
| DQL/ Data Practice Group 1, Biomedical Data<br>Sciences Department, Japan | 14-SEP-2018 | eSignature |
| PPD OSL/ Clinical Operation Department, Japan | 13-SEP-2018 | eSignature |
| PPD Lead programmer/ Manager, Statistical | 18-SEP-2018 | eSignature |
| Programming & Reporting Group, Biomedical Data Sciences Department, Japan | 10-021-2010 | corgnature |
| Clinical Scientist/ Respiratory TA Office,<br>Medicines Development, Japan | 13-SEP-2018 | eSignature |
| SAP/CIL/ Infectious Disease/ Future Pipelines Discovery Office, Medicines Development, Japan | 13-SEP-2018 | eSignature |
| Medical Writing/ Manager, Medical Writing Office, Medicines Development, Japan | 13-SEP-2018 | eSignature |
| Medical Lead/ Manager, MA Immuno-<br>Inflammation & Infectious Disease Department,<br>Japan | 13-SEP-2018 | eSignature |
| Clinical Safety Expert/ PV Information Management Service Department., Japan | 13-SEP-2018 | eSignature |

## The GlaxoSmithKline group of companies

# Clinical Statistics and Clinical Programming Line Approvals: Approved by (Approvals captured electronically in CARS system):

| Approver | Date | Approval Method |
|---|---|---|
| PPD | | |
| Clinical Statistics Line Approver/ Manager,<br>Biostatistics Group 1, Biomedical Data Sciences<br>Department, Japan. | 18-SEP-2018 | eSignature |
| PPD | | |
| Clinical Programming Line Approver / Department Manager, Biomedical Data Sciences Department, Japan. | 18-SEP-2018 | eSignature |

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTR | ODUCTION | 7 |
| 2. | SUMI | MARY OF KEY PROTOCOL INFORMATION | 7 |
| | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | |
| 3. | PLAN | NED ANALYSES | 9 |
| | 3.1. | Interim Analyses | |
| | 3.2. | Primary Analyses (WEEK 48) | |
| | 3.3. | Final Analyses (WEEK 96) | 9 |
| 4. | | YSIS POPULATIONS | |
| | 4.1. | Protocol Deviations | |
| | 4.2. | Efficacy Evaluable Set | 10 |
| 5. | CON | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | VENTIONS | |
| | 5.1. | Study Treatment & Subgroup Display Descriptors | |
| | 5.2. | Baseline Definitions | 11 |
| | 5.3. | Examination of Covariates, Other Strata and Subgroups | |
| | <b>5</b> 4 | 5.3.1. Examination of Subgroups | |
| | 5.4. | Multiple Comparisons and Multiplicity | 12 |
| | 5.5. | Other Considerations for Data Analyses and Data Handling Conventions | 13 |
| _ | OTLIF | DV DODULATION ANALYOFO | 4.4 |
| 6. | 6.1. | OY POPULATION ANALYSES | |
| | 0.1. | Overview of Planned Study Population Analyses | 14 |
| 7. | EFFI( | CACY ANALYSES | |
| | 7.1. | Primary Efficacy Analyses | |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | |
| | | 7.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.1.5. Statistical Analyses / Methods | 15 |
| | | 7.1.5.1. Overview of Planned Efficacy Analyses | |
| | 7.2. | 3, 1, 1 | |
| | 1.2. | Secondary Efficacy Analyses7.2.1. Endpoint / Variables | |
| | | 7.2.2. Summary Measure | |
| | | 7.2.3. Population of Interest | |
| | | 7.2.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.2.5. Statistical Analyses / Methods | |
| | | 7.2.5.1. Overview of Planned Efficacy Analyses | |
| | | 7.2.5.2. Statistical Methodology Specification | |


| 8. | SAFET | TY ANALYSES | 21 |
|---|---|---|---|
| | 8.1. | Adverse Events Analyses | 21 |
| | 8.2. | Adverse Events of Special Interest Analyses | |
| | 8.3. | Clinical Laboratory Analyses | |
| | 8.4. | Other Safety Analyses | 23 |
| 9. | EXPLO | ORATORY EFFICACY ANALYSES | 25 |
| | 9.1. | HBsAg Responder/Non-Responder Analyses | |
| | 9.2. | ALT Categories Analyses | 26 |
| | 9.3. | Correlation of virus parameters | 28 |
| | 9.4. | Background factor of HBsAg Responder/ Non-Responder | 28 |
| | 9.5. | Safety Subgroup Analysis | |
| 10. | REFE | RENCES | 30 |
| 11 | APPEN | NDICES | 31 |
| • • • | 11.1. | | |
| | | 11.1.1. Exclusions from Efficacy Evaluable Set | |
| | 11.2. | Appendix 2: Schedule of Activities | 32 |
| | | 11.2.1. Protocol Defined Schedule of Events | |
| | 11.3. | Appendix 3: Assessment Windows | |
| | | 11.3.1. Definitions of Assessment Windows for Analyses | |
| | | 11.3.2. Selection of Data in the Event of Multiple Records in a | |
| | | Window11.3.2.1. Serology, ALT and Laboratory Parameters of | 36 |
| | | Interest | 36 |
| | | 11.3.2.2. HBV DNA values (log10 IU/mL) | 37 |
| | 11.4. | 11 | |
| | | 11.4.1. Study Phases | |
| | | 11.4.1.1. Study Phases for Concomitant Medication | |
| | | 11.4.2. Treatment States for AE data | |
| | 11.5. | Appendix 5: Data Display Standards & Handling Conventions | |
| | | 11.5.1. Reporting Process | |
| | 44.0 | 11.5.2. Reporting Standards | |
| | 11.6. | | |
| | | 11.6.1. General | |
| | | 11.6.2. Study Population | |
| | | 11.6.3. Efficacy | |
| | 11.7. | 11.6.4. Safety Appendix 7: Reporting Standards for Missing Data | |
| | 11.7. | 11.7.1. Premature Withdrawals | |
| | | 11.7.2. Handling of Missing Data | |
| | | 11.7.2.1. Handling of Missing and Partial Dates | |
| | | 11.7.2.2. Handling of Missing Data for Statistical | 41 |
| | | Analysis | 48 |
| | 11.8. | | 40 |
| | | 11.8.1. LDTA GSI grading scale (LDTA GSI grade) | |
| | | 11.8.2. GSI modified NIAID Common Toxicity Grading Scale (GSI | |
| | | NIAID grade) | 52 |
| | 11.9. | | |
| | | Appendix 10: Viread (Tenofovir Disoproxil Fumarate) Risk | |
| | | Management Plan for the ELL (Version 22) January 2017 | 57 |


| 11.11. | Appendix | ( 11: Abbreviations & Trade Marks | 59 |
|--------|-------------|---------------------------------------------|----|
| | 11.11.1. | Abbreviations | 59 |
| | 11.11.2. | Trademarks | 59 |
| 11.12. | | c 12: List of Data Displays | |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverables | |
| | | Study Population Tables | |
| | | Efficacy Tables | |
| | | Efficacy Figures | |
| | | Safety Tables | |
| | | Safety Figures | |
| | | Exploratory Statistical Analysis Tables | |
| | | Exploratory Statistical Analysis Figures | |
| | | ICH Listings | |
| 11 13 | | x 13: Example Mock Shells for Data Displays | |
| 11.10. | , wpcilluis | t to. Example wook offers for bala bisplays | -0 |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:205883.

| Revision Chronolog | y: | |
|--------------------|-------------|----------|
| Ver. 0 | 18-SEP-2018 | Original |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 6 (Dated: 5/JUL/2018).

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the HBsAg | • Proportion of subjects achieving 0.25 Log <sub>10</sub> |
| reduction potential at week 48 | HBsAg reduction from the baseline at week 48 |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the virological | • Proportion of subjects achieving 0.25 Log <sub>10</sub> |
| effects | HBsAg reduction from the baseline at week 24 |
| | and 96 |
| | Proportion of subjects achieving HBsAg loss |
| | and HBsAg/Ab seroconversion at week 24, 48 |
| | and 96 |
| | Proportion of subjects achieving HBeAg loss |
| | and HBeAg/Ab seroconversion at week 24, 48 |
| | and 96 |
| | • Reduction of HBsAg titer from the baseline at |
| | week 24, 48 and 96 |
| | • Reduction of HBcrAg titer from the baseline at |
| | week 24, 48 and 96 |
| Safety | Safety Endpoints |
| To evaluate Safety | • AE |
| | Clinical laboratory values |
| | Vital signs |
| | • ECG |
| | Bone density |

## 2.3. Study Design



# 2.4. Statistical Hypotheses / Statistical Analyses

No formal statistical hypotheses will be tested. Descriptive statistics will be used to assess the efficacy and safety objectives. An estimation approach will be used to address the efficacy objectives, where point estimates and corresponding 95% confidence intervals will be constructed.

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

Interim analysis to make statistical investigations will not be performed in this study.

## 3.2. Primary Analyses (WEEK 48)

The CRF data by Week 48 will be locked when all subjects (excluding withdrawn subjects) complete Week48 to collect safety and efficacy data. Safety and efficacy data will be analysed after the completion of all required database cleaning activities have been completed and database release (DBR) and Data Base Freeze (DBF) has been declared by Data Management.

Even though this is a single arm study, randomisation codes will be distributed according to RandAll NG procedures.

## 3.3. Final Analyses (WEEK 96)

Week 96 planned analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final DBR and DBF has been declared by Data Management.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | <b>Analyses Evaluated</b> |
|---|---|---|
| Enrolled | Subjects who provided consent | Study Population |
| Screening<br>Failure | Subjects who provided consent but were not subsequently administered. | Study Population |
| Safety<br>Population (SP) | Subjects who have received at least one dose of study treatment after enrolment. | • Safety |
| Full Analysis<br>Set (FAS) | A population of all subjects enrolled in the study, excluding those who meet either of the following criteria: | • Efficacy |
| | <ul> <li>Have not received any dose of study treatment.</li> </ul> | |
| | <ul> <li>Have no efficacy data* (HBsAg, HBV-DNA,<br/>HBcrAg, HBeAg, HBsAb, HBeAb, ALT)<br/>after the start of study treatment.</li> </ul> | |
| | *: at least 15 days after the start of study treatment. | |
| Efficacy<br>Evaluable Set<br>(EES) | A subset of subjects in the FAS defined above and evaluable for efficacy. | • Efficacy |

Refer to Appendix 12 List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

• Data will be reviewed prior to freezing the database to ensure all important deviations. This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

## 4.2. Efficacy Evaluable Set

Details of efficacy evaluable set will be provided in Section 11.1.1.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Subgroup Display Descriptors

| Treatment Group Descriptions | | | | |
|---|---|---|---|---|
| RandAll NG | RandAll NG Data Displays for Reporting | | | |
| Code | Descripti | ion | Description | Order in TLF |
| T | T | | TDF | 1 |

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | Study Assessments Considered as Baseline | | Baseline Used in Data<br>Display |
|---|---|---|---|
| | Screening | Day 1 (Pre-<br>Dose) | |
| Efficacy | | | |
| HBV-DNA | X | X | Day1 |
| ALT | X | X | Day1 |
| HBeAg/Anti-HBe | X | X | Day1 |
| HBsAg/Anti-HBs | X | X | Day1 |
| HBcrAg | | X | Day1 |
| Safety | | | |
| 12 Lead ECG | X | | Screening |
| Vital Signs | X | X | Day 1 |
| Haematology | X | X | Day 1 |
| Clinical Chemistry | X | X | Day 1 |
| Urine Analysis | X | X | Day 1 |
| Bone density (absolute) | X | | Screening |

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing. Note that height and weight in screening will be used for demographic characteristics.

## 5.3. Examination of Covariates, Other Strata and Subgroups

#### 5.3.1. Examination of Subgroups

The list of subgroups may be used in descriptive summaries. Additional subgroups of clinical interest may also be considered.

| Subgroup | Categories |
|---|---|
| Protocol defined liver | Yes, No |
| cirrhosis | |
| Genotype | A, B, C, D |
| HBsAg subgroup category | <800 KIU/L, >=800 KIU/L |
| HBsAg subgroup category (Conventional unit) | <800 IU/mL, >=800 IU/mL |
| AGE category | <40, 40-49, 50-59, 60- |
| Former Peg-INF (within 2 | Yes, No |
| years prior to screening) | Note: Peg-Interferon codes are listed in Appendix 9. |

## **Exploratory Analysis**

| Subgroup | Categories |
|---|---|
| HBsAg responder / Non-<br>responder at WEEK 48 | <= -0.25 log10 HBsAg, > -0.25 log10 HBsAg |
| ALT category*1 | <60 IU/L, >=60 IU/L |
| ALT category* <sup>2</sup> (Conventional unit) | <60 U/L, >=60 U/L |

#### **NOTES:**

- \*1: >=60 IU/L of ALT category is 60 or more than 60 from baseline to WEEK 48 <60 IU/L of ALT category is less than 60 from baseline to WEEK 48
- \*2: >=60 U/L of ALT category is 60 or more than 60 from baseline to WEEK 48 <60 U/L of ALT category is less than 60 from baseline to WEEK 48

## Safety Subgroup Analysis

| Subgroup | Categories |
|---|---|
| AGE category | <40, 40-49, 50-59, 60- |
| eGFR (ml/sec/1.73m <sup>2</sup> ) baseline category | <1, 1<= - <1.5, >=1.5 |
| eGFR (ml/min/1.73m²)<br>baseline category<br>(Conventional unit) | <60, 60<= - <90, >=90 |
| Weight baseline category | <50 kg, >=50 kg |
| Sex | Male, Female |

# 5.4. Multiple Comparisons and Multiplicity

Analyses of efficacy endpoints will not be subject to any multiplicity adjustment.

# 5.5. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| 11.3 | Appendix 3: Assessment Windows |
| 11.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 11.6 | Appendix 6: Derived and Transformed Data |
| 11.7 | Appendix 7: Reporting Standards for Missing Data |
| 11.8 | Appendix 8: Values of Potential Clinical Importance |
| 11.9 | Appendix 9 Listing of Peg-Interferon codes |
| 11.10 | Appendix 10 Viread (Tenofovir Disoproxil Fumarate) Risk Management Plan for the EU |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "Safety" or "FAS" or "EES" population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 12: List of Data Displays.

Other baseline characteristics, e.g. virus characteristics (Screening: Genotype, Baseline: Serum HBV-DNA, Serum ALT, HBeAg, HBsAg, HBcrAg), Prior medical condition and Protocol defined liver cirrhosis will be summarized. To check baseline values for HBsAg, HBcrAg, ALT and HBV-DNA, summary statistics at baseline will be shown.

#### **Overview of Planned Study Population Analyses**

| [Endpoint / Parameter / Display Type] | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| <b>Subject Disposition</b> | | | |
| Subject Disposition and Reason for Study<br>Withdrawal | Y | | Y |
| Screening Status and Reasons for Screen Failure | Y | | Y |
| <b>Protocol Deviations</b> | • | | |
| Important Protocol Deviations | Y | | Y |
| Subjects with Inclusion/Exclusion Criteria<br>Deviations | Y | | Y |
| Populations Analysed | • | | |
| Study Populations | Y | | |
| Subjects Excluded from EES Population | | | Y |
| <b>Demographic and Baseline Characteristics</b> | • | | |
| Demographic Characteristics | Y | | Y |
| Demographic Characteristics for Screening Failure | Y | | Y |
| Age Ranges | Y | | |
| Race and Racial Combinations | Y | | Y |
| Other Baseline Characteristics | Y | | Y |
| <b>Medical Conditions and Concomitant Medications</b> | | | |
| Medical Conditions | Y | | Y |
| Prior Hepatitis Medications | Y | | Y |
| Concomitant Medications | Y | | Y |
| <b>Exposure and Treatment Compliance</b> | | | |
| Exposure to Study Treatment | Y | | Y |
| Treatment Compliance | Y | | Y |
| Subgroup | | | |
| Demographic Characteristics | Y | | |

**NOTES:** Y = Yes display generated.

#### 7. EFFICACY ANALYSES

## 7.1. Primary Efficacy Analyses

### 7.1.1. Endpoint / Variables

HBsAg responder proportion of subjects with -0.25 or less log<sub>10</sub> HBsAg change from baseline switching from Entecavir to Tenofovir at Week 48.

## 7.1.2. Summary Measure

Proportion of HBsAg responder subjects with -0.25 or less log<sub>10</sub> HBsAg change from baseline switching from Entecavir to Tenofovir at Week 48.

## 7.1.3. Population of Interest

The primary efficacy analyses will be based on the "FAS" population. Also "EES" population will be applied to investigate the robustness of the primary result.

#### 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

If any subjects will be discontinued due to AE or rescue medication before Week 48, data collection at Week 48 will not be conducted. However, in order to evaluate primary endpoint at Week 48, any subjects withdrawn from the study will be treated as non-responders (defined as subjects not achieving 0.25 log<sub>10</sub> HBsAg reduction from the baseline at Week 48).

## 7.1.5. Statistical Analyses / Methods

#### 7.1.5.1. Overview of Planned Efficacy Analyses

| [Endpoint / | Absolute | | | | | | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | Stats | | Summar | | Indi | Individu | | Stats | | | Summar | | Individu | |
| Type] | Analysis | | 3 | y | | al | | Analysis | | | y | | al | |
| | T | F | L | T | F | F | L | T | F | L | T | F | F | L |
| HBsAg | | | | | | | | | | | | | | |
| HBsAg responder | | | | Y | | | | | | | | | | |
| proportion | | | | | | | | | | | | | | |
| (WEEK 48) | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data
- Individual = Represents FL related to any displays of individual subject observed raw data.

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, and listed.

#### 7.1.5.2. Statistical Methodology Specification

#### **Endpoint / Variables**

• HBsAg responder proportion of subjects with -0.25 or less log<sub>10</sub> HBsAg change from baseline switching from Entecavir to Tenofovir at week 48.

#### **Model Specification**

• N/A

#### **Model Checking & Diagnostics**

N/A

#### **Model Results Presentation**

N/A

#### **Subgroup Analyses**

• The analysis on the primary endpoint will be also performed for subgroups. Subgroup analyses are intended to confirm the robustness of results. Refer to Section 5.3.1.

## **Sensitivity and Supportive Analyses**

• Supportive Analysis: "EES" population will be applied to investigate the robustness of the primary result.

## 7.2. Secondary Efficacy Analyses

#### 7.2.1. Endpoint / Variables

Refer to "Endpoint / Variables and Summary Measure" in Section 7.2.5.2.

#### 7.2.2. Summary Measure

Refer to "Endpoint / Variables and Summary Measure" in Section 7.2.5.2.

#### 7.2.3. Population of Interest

The secondary efficacy analyses will be based on the "FAS" or "EES" population, unless otherwise specified.

#### 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

For binomial variables, the strategy for intercurrent events will be according to Section 7.1.4. For continuous variables, if subjects will be withdrawn from the study due to adverse events or rescue medication before Week 48/Week 96, data after withdrawal

will not be collected, and data analysis will be performed on collected data (i.e. After withdrawal, data will not be collected and data will not be imputed.).

## 7.2.5. Statistical Analyses / Methods

## 7.2.5.1. Overview of Planned Efficacy Analyses

| [Endpoint / | Absolute | | | | | | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ | | Stats | | Sum | mar | Indi | vidu | | Stats | | | ımar | | vidu | |
| Display Type] | A | nalys | is | у | | a | .1 | Analysis | | | | у | | а | .1 |
| | T | F | L | Т | F | F | L | T | F | L | Т | F | F | L | |
| HBsAg | | | | | | | | | | | | | | | |
| Frequency of | | | | Y | | | Y | | | | | | | | |
| HBsAg responder | | | | | | | | | | | | | | | |
| Proportion | | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | | |
| Summary of log <sub>10</sub> | | | | Y | Y | | Y | | | | Y | Y | | Y | |
| HBsAg | | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | | |
| Summary of | | | | Y | | | Y | | | | Y | | | Y | |
| HBsAg | | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | | |
| Frequency of | | | | Y | | | | | | | | | | | |
| HBsAg category | | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | | |
| Summary of log <sub>10</sub> | | | | Y | Y | | Y | | | | Y | Y | | Y | |
| HBsAg with | | | | | | | | | | | | | | | |
| conventional unit | | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | | |
| Summary of | | | | Y | | | Y | | | | Y | | | Y | |
| HBsAg with | | | | | | | | | | | | | | | |
| conventional unit | | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | | |
| Frequency of | | | | Y | | | | | - | | | | | | |
| HBsAg category | | | | | | | | | | | | | | | |
| with conventional | | | | | | | | | | | | | | | |
| unit (Study visit up | | | | | | | | | | | | | | | |
| to 48/96 weeks) | | | | | | | | | | | | | | | |
| Seroconversion | | | | | | | | | | | | | | | |
| Proportion of | | | | Y | | | Y | | - | | | | | | |
| subjects achieving | | | | | | | | | | | | | | | |
| HBsAg loss | | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | | |
| Proportion of | | | | Y | | | Y | | | | | | | | |

| [Endpoint / | Absolute Change from Ba | | | | | | | | Base | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ | | Stats | | Sum | | Indi | vidu | | Stats | | | ımar | | vidu |
| Display Type] | Α | nalys | is | 7 | | a | | <i>A</i> | Analys | | | <b>V</b> | а | |
| I A Alexander | T | F | L | T | F | F | L | T | F | L | Т | F | F | L |
| subjects achieving | | | | | | | | | | | | | | |
| HBsAg/Ab | | | | | | | | | | | | | | |
| seroconversion a | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Proportion of | | | | Y | | | Y | | | | | | | |
| subjects achieving | | | | 1 | | | • | | | | | | | |
| HBeAg loss | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Proportion of | | | | Y | | | Y | | | | | | | |
| subjects achieving | | | | 1 | | | 1 | | | | | | | |
| HBeAg/Ab | | | | | | | | | | | | | | |
| seroconversion | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | <u> </u> | <u> </u> | <u> </u> | | | | | | | | | |
| Virology | I | 1 | 1 | 17 | 17 | | 17 | l | I | I | 17 | 17 | | 37 |
| Summary of | | | | Y | Y | | Y | | | | Y | Y | | Y |
| HBcrAg | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Frequency of | | | | Y | | | | | | | | | | |
| HBcrAg category | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Summary of HBV- | | | | Y | Y | | Y | | | | Y | Y | | Y |
| DNA (Study visit | | | | | | | | | | | | | | |
| up to 48/96 weeks) | | | | | | | | | | | | | | |
| Summary of | | | | Y | | | Y | | | | Y | | | Y |
| HBeAg | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Summary ofLog <sub>10</sub> | | | İ | Y | İ | | Y | | | | Y | Y | | Y |
| HBeAg | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Frequency of | | İ | t | Y | t | | Y | | | | | | | |
| Virological | | | | | | | 1 | | | | | | | |
| Breakthrough | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Summary of | | | | Y | Y | | Y | | | | Y | Y | | Y |
| HBcrAg with | | | | 1 | 1 | | 1 | | | | 1 | 1 | | 1 |
| conventional unit | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | <u> </u> | 17 | | | | | | | | | | |
| Frequency of | | | | Y | | | | | | | | | | |
| HBcrAg category | | | | | | | | | | | | | | |

| [Endpoint / | | Absolute | | | | | | | Ch | ange | from | Base | line | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ | | Stats | | Sum | mar | Indi | vidu | | Stats | | Sum | ımar | Indi | vidu |
| Display Type] | A | nalys | is | 3 | 7 | a | al | | alys | sis | У | | al | |
| | T | F | L | T | F | F | L | T | F | L | T | F | F | L |
| with conventional | | | | | | | | | | | | | | |
| unit | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| ALT | | | | | | | | | | | | | | |
| Summary of ALT | | | | Y | Y | | Y | | | | Y | Y | | Y |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Summary of ALT | | | | Y | Y | | Y | | | | Y | Y | | Y |
| with conventional | | | | | | | | | | | | | | |
| unit | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |

#### **NOTES:**

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- HBV-DNA: Source data is log<sub>10</sub> IU/mL.
- HBcrAg: Source data is log<sub>10</sub> IU/mL
- Up to 48 weeks: Baseline, 4, 12, 24, 36, 48 week
- UP to 96 weeks: Baseline,4,12,24,36,48,60,72,84,96 week

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.2.5.2. Statistical Methodology Specification

#### **Endpoint / Variables and Summary Measures**

- Proportion of HBsAg responder subjects with -0.25 or less log<sub>10</sub> HBsAg change from baseline switching from Entecavir to Tenofovir (HBsAg responder) up to week 48 /week96
- Summary of log<sub>10</sub> HBsAg up to week 48/ week 96 including change from baseline
- Summary of HBsAg up to week 48/ week 96 including change from baseline
- Frequency of HBsAg category up to week 48/ week 96
- Summary of HBV-DNA up to week 48/ week 96 including change from baseline
- Summary of HBcrAg up to week 48/ week 96 including change from baseline
- Frequency of HBcrAg category up to week 48/ week 96

- Summary of ALT up to week 48/ week 96 including change from baseline
- Proportion of subjects achieving HBsAg loss up to week 48/ week 96
- Proportion of subjects achieving HBsAg/Ab seroconversion up to week 48/ week 96
- Proportion of subjects achieving HBeAg loss up to week 48/ week 96
- Proportion of subjects achieving HBeAg/Ab seroconversion up to week 48/ week 96
- Summary of HBeAg up to week 48/ week 96 including change from baseline
- Summary of log<sub>10</sub> HBeAg up to week 48/ week 96 including change from baseline
- Proportion of subjects achieving Virological Breakthrough (Week 0 -Week 48 /Week 96)
- Summary of log<sub>10</sub> HBsAg (conventional unit) up to week 48/ week 96 including change from baseline
- Summary of HBsAg (conventional unit) up to week 48/ week 96 including change from baseline
- Frequency of HBsAg category (conventional unit) up to week 48/ week 96
- Summary of HBcrAg (conventional unit) up to week 48/ week 96 including change from baseline
- Frequency of HBcrAg category (conventional unit) up to week 48/ week 96
- Summary of ALT (conventional unit) up to week 48/ week 96 including change from baseline

#### **Model Specification**

N/A

#### **Model Checking & Diagnostics**

N/A

#### **Model Results Presentation**

N/A

#### **Subgroup Analyses**

- The analysis on the secondary endpoint (log<sub>10</sub> HBsAg, HBcrAg\*, log<sub>10</sub> HBeAg) will be also performed for subgroups. These subgroup analyses are intended to confirm the robustness of results. Refer to Section 5.3.1.
  - \*: Source data is log<sub>10</sub>

#### **Sensitivity and Supportive Analyses**

• Supportive Analysis: "EES" population will be applied to investigate the robustness of the primary result (HBsAg responder proportional Week 48).

#### 8. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, unless otherwise specified.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious adverse events (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 12: List of Data Displays.

## 8.2. Adverse Events of Special Interest Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event (See the list of Adverse Event of special interest in Section 11.6.4.). Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be re-reviewed by the Medical Monitor in place at the time of reporting.

The details of the planned displays are provided in Appendix 12: List of Data Displays.

#### **Overview of Planned Adverse Event Analyses**

| Display Type | | Absolu | lute |
|---|---|---|---|
| | Sum | mary | Individu |
| | | | al |
| | T | F | L |
| Adverse Events (AEs) | | | |
| All AEs by SOC and PT | Y | | Y |
| All AEs by Maximum Intensity | Y | | |
| Drug-Related AEs by SOC and PT | Y | | |
| Drug-Related AEs by Maximum Intensity | Y | | |
| Subject Numbers for Individual AEs | | | Y |
| Relationship Between AE SOCs, PT and Verbatim Text | | | Y |
| Serious AEs | | | |
| All Serious AEs | Y | | Y |
| Fatal Serious AEs | Y | | Y |
| Other Significant AEs | | | |
| AEs Leading to Withdrawal from Study | Y | | Y |
| AE of special interest | | | |
| Renal AE | Y | | Y |
| Bone Events | Y | | Y |
| Liver AE | Y | | Y |

#### NOTES:

• T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred Term.

- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 12: List of Data Displays.

## **Overview of Planned Clinical Laboratory Analyses**

| Display Type | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | | nmar<br>y | Individu<br>al | Sum | mary | Indiv<br>idual |
| | T | F | L | T | F | L |
| Chemistry | | | | | | |
| Chemistry Data | Y | | Y | Y | | Y |
| Chemistry Results Relative to Normal Range | | | | Y | | |
| Creatinine | | Y | | | Y | |
| eGFR | | Y | | | Y | |
| Corrected calcium based on the serum albumin | Y | | Y | | | |
| Chemistry (ALT, ALP, Creatinine, Phosphorus, Glucose, Uric acid, eGFR) Data with conventional unit | Y | | Y | Y | | Y |
| Creatinine with conventional unit | | Y | | | Y | |
| eGFR with conventional unit | | Y | | | Y | |
| Hematology | | | | | | |
| Hematology Data | Y | | Y | Y | | Y |
| Hematology Results Relative to Normal Range | | | | Y | | |
| Urinalysis | | | | | | |
| Glucose, protein, urinary sediment | Y | | Y | | | |
| β2-microglobulin, β2-microglobulin-creatinine ratio, %TRP creatinine, electrolyte (P) | Y | | Y | Y | | Y |
| Urinalisis (β2-microglobulin, electrolyte (P),<br>Creatinine) with conventional unit | Y | | Y | Y | | Y |
| Hepatobiliary (Liver) <sup>[1]</sup> | | | | | | |
| Liver Monitoring/Stopping Event Reporting | Y | | Y | | | |
| Medical Conditions for Subjects with Liver<br>Stopping Events | Y | | Y | | | |
| Substance Use for Subjects with Liver Stopping Events | Y | | Y | | | |
| LDTA GSI grade scale | | | | | | |
| Treatment-Emergent Laboratory Abnormalities, | Y | | Y | | | |

| Display Type | | Abso | olute | Chai | nge fror | n BL |
|---|---|---|---|---|---|---|
| | Sum | mar | Individu<br>al | Sum | mary | Indiv<br>idual |
| | T | F | L | T | F | L |
| LDTA GSI grading scale | | | | | | |
| LDTA GSI Grade 3/4 Treatment-Emergent<br>Laboratory Abnormalities | Y | | Y | | | |
| Treatment-Emergent Marked Laboratory<br>Abnormalities, LDTA GSI grading scale | Y | | Y | | | |
| Hepatic Flare | _ | | | | | |
| On-Treatment Hepatic Flare | Y | | Y | | | |
| On-Treatment Laboratory Values Relevant to on-<br>Treatment Hepatic Flare | Y | | Y | | | |
| Renal Parameters | _ | | | | | |
| Confirmed Changes in Renal Parameters | Y | | Y | | | Y |
| GSI Modified NIAID | _ | | | | | |
| Treatment-Emergent Laboratory Abnormalities,<br>GSI Modified NIAID | Y | | Y | | | |
| GSI Modified NIAID Grade 3/4 Treatment-<br>Emergent Laboratory Abnormalities | Y | | Y | | | |
| Treatment-Emergent Marked Laboratory<br>Abnormalities, GSI Modified NIAID | Y | | Y | | | |

#### **NOTES:**

- T = Table, F = Figures, L = Listings, Y = Yes display generated
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 12: List of Data Displays.

#### **Overview of Planned Other Safety Analyses**

| Display Type | Absolute | | olute | Cha | nge fr | om BL |
|---|---|---|---|---|---|---|
| | Summar<br>y | | Individu<br>al | Sum | mary | Indivi<br>dual |
| | T | F | L | T | F | L |
| ECG | | | | | | |
| ECG Findings | Y | | Y | | | |

<sup>&</sup>lt;sup>1</sup>: If Hepatobiliary will be occurred.

| Display Type | | Abso | olute | Cha | nge fr | om BL |
|---|---|---|---|---|---|---|
| | Sum | ımar<br>Y | Individu<br>al | Sum | mary | Indivi<br>dual |
| | T | F | L | T | F | L |
| ECG Values | Y | | Y | Y | | Y |
| Vital Signs | | | | | | |
| Vitals Values | Y | | Y | Y | | Y |
| Others | | | | | | |
| Bone density (%)* | | | | Y | Y | Y |
| Bone density (absolute) | Y | | Y | Y | Y | Y |

#### **NOTES:**

- T = Table, F = Figures, L = Listings, Y = Yes display generated
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- \*:Bone density (%): %change from baseline
- Bone density data: DEXA method will be displayed by position

## 9. EXPLORATORY EFFICACY ANALYSES

## 9.1. HBsAg Responder/Non-Responder Analyses

Summary statistics of efficacy parameter by HBsAg responder/Non-responder at WEEK 48 will be provided Frequency of HBsAg responder/Non-responder with ALT category (<60 IU/L, >=60 IU/L) and with ALT category (<60 U/L, >=60 U/L; conventional unit) at WEEK 48 will be provided (Cross Table).

Listing of subject numbers for individual HBsAg Responder/Non-Responder Category at WEEK 48 will be provided.

These analyses will be based on the "FAS" population, unless otherwise specified. The details of the planned displays are presented in Appendix 12: List of Data Displays.

## **Overview of Planned Exploratory Efficacy Analyses**

| [Endpoint / | | | | Abso | olute | | | | ( | Chan | ge fro | m Ba | seline | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | 5 | Stats | 5 | Sum | mary | Indiv | ridual | | Stat | S | Sum | mary | Indiv | ridual |
| Type] | Ar | nalys | sis | | | | | Aı | naly | sis | | - | | |
| | T | F | L | T | F | F | L | T | F | L | T | F | F | L |
| HBsAg | | | | | | | | | | | | | | |
| Summary of log <sub>10</sub> | | | | Y | Y | | | | | | Y | Y | Y | |
| HBsAg | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Summary of log <sub>10</sub> | | | | Y | Y | | | | | | Y | Y | Y | |
| HBsAg with | | | | | | | | | | | | | | |
| conventional unit | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Other Efficacy | 1 | ı | ı | | ** | 1 | I | | ı | 1 | ** | ** | | I |
| Summary of HBcrAg | | | | Y | Y | | | | | | Y | Y | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | 3.7 | 3.7 | | | | | | Y | 3.7 | | |
| Summary of HBV- | | | | Y | Y | | | | | | Y | Y | | |
| DNA (Study visit up | | | | | | | | | | | | | | |
| to 48/96 weeks) | | | | Y | Y | | | | | | Y | Y | | |
| Summary of ALT (Study visit up to | | | | Y | Y | | | | | | Y | Y | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Summary of log <sub>10</sub> | | | | Y | Y | | | | | | Y | Y | | |
| HBeAg | | | | 1 | 1 | | | | | | 1 | 1 | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Other Efficacy (Conve | ntio | nal ı | ınit | ) | | | <u> </u> | | | | <u> </u> | <u> </u> | | <u> </u> |
| Summary of HBcrAg | | | | Y | Y | | | | | | Y | Y | | |
| with conventional unit | | | | | | | | | | | _ | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Summary of ALT | | | | Y | Y | | | | | | Y | Y | | |

| [Endpoint / | | Absolute | | | | | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | 5 | Stats | | Sumi | mary | Indiv | idual | | Stats | S | Sum | mary | Indiv | idual |
| Type] | Ar | alys | sis | | | | | A | naly | sis | | - | | |
| | T | F | L | T | F | F | L | T | F | L | T | F | F | L |
| with conventional unit<br>(Study visit up to<br>48/96 weeks) | | | | | | | | | | | | | | |

#### **NOTES:**

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Subject's number for individual HBsAg Responder/Non-Responder category at WEEK 48 will be listed
- Up to 48 weeks: Baseline, 4, 12, 24, 36, 48 week
- UP to 96 weeks: Baseline, 4, 12, 24, 36, 48, 60, 72, 84, 96 week

## 9.2. ALT Categories Analyses

Summary statistics of efficacy parameter by ALT category (<60 IU/L, >=60 IU/L) at WEEK 48 will be provided.

Summary statistics of efficacy parameter (Conventional unit) by ALT category with conventional unit (<60 U/L, >=60 U/L) at WEEK 48 will be provided.

Listing of subject numbers for individual ALT Category (<60 IU/L, >=60 IU/L) at WEEK 48 will be provided.

Listing of subject numbers for individual ALT Category with conventional unit (<60 U/L, >=60 U/L) at WEEK 48 will be provided.

These analyses will be based on the "FAS" population, unless otherwise specified. The details of the planned displays are presented in Appendix 12: List of Data Displays.

#### **Overview of Planned Exploratory Efficacy Analyses**

| [Endpoint / | | Absolute | | | | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | , | Stats | | Sumi | mary | Indiv | idual | | Stats | S | Sum | mary | Indiv | ridual |
| Type] | Aı | nalys | sis | | | | | A | nalys | sis | | | | |
| | T | F | L | T | F | F | L | T | F | L | T | F | F | L |
| HBsAg | | | | | | | | | | | | | | |
| Summary of log <sub>10</sub> | | | | Y | Y | | | | | | Y | Y | | |
| HBsAg | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| HBsAg with convention | HBsAg with conventional unit ALT category (<60 U/L, >=60 U/L) | | | | | | | | | | | | | |
| Summary of log <sub>10</sub> | | | | Y | Y | | | | | | Y | Y | | |

| [Endpoint / | | | | Abso | lute | | | | ( | Chan | ge fro | m Bas | seline | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | , | Stats | ; | Sum | mary | Indiv | ridual | | Stats | | | mary | | ridual |
| Type] | Aı | nalys | sis | | • | | | Α | naly | sis | | , | | |
| | T | F | L | T | F | F | L | T | F | L | T | F | F | L |
| HBsAg with | | | | | | | | | | | | | | |
| conventional unit | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Other Efficacy | | | | | | | | | | | | | | |
| Summary of HBcrAg | | | | Y | Y | | | | | | Y | Y | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Summary of HBV- | | | | Y | Y | | | | | | Y | Y | | |
| DNA (Study visit up | | | | | | | | | | | | | | |
| to 48/96 weeks) | | | | | | | | | | | | | | |
| Summary of ALT | | | | Y | Y | | | | | | Y | Y | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Summary of log <sub>10</sub> | | | | Y | Y | | | | | | Y | Y | | |
| HBeAg | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |
| Other Efficacy with co | onve | ntio | nal | | 1 | ategor | y (<60 | U/I | ۰, >= | 60 U | | 1 | 1 | 1 |
| Summary of HBcrAg | | | | Y | Y | | | | | | Y | Y | | |
| with conventional | | | | | | | | | | | | | | |
| unit (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | L | | | | | | | | | | |
| Summary of HBV- | | | | Y | Y | | | | | | Y | Y | | |
| DNA (Study visit up | | | | | | | | | | | | | | |
| to 48/96 weeks) | | | | | | | | | | | | | | |
| Summary of ALT | | | | Y | Y | | | | | | Y | Y | | |
| with conventional | | | | | | | | | | | | | | |
| unit (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | 177 | * 7 7 | | | | | | 17 | 7.7 | | |
| Summary of log <sub>10</sub> | | | | Y | Y | | | | | | Y | Y | | |
| HBeAg | | | | | | | | | | | | | | |
| (Study visit up to | | | | | | | | | | | | | | |
| 48/96 weeks) | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Subject's number for individual ALT category (<60 IU/L, >=60 IU/L) at WEEK 48 will be listed.

## 9.3. Correlation of virus parameters

These analyses will be based on the "FAS" population, unless otherwise specified.

Following correlation plots will be provided.

- log<sub>10</sub> HBsAg change from baseline vs ALT change from baseline (WEEK24/WEEK48/ WEEK96)
- log<sub>10</sub> HBsAg change from baseline vs HBcrAg baseline (WEEK24/WEEK48/WEEK96)
- log<sub>10</sub>HBsAg change from baseline vs HBcrAg change from baseline (WEEK24/WEEK48/WEEK96)
- log<sub>10</sub>HBsAg change from baseline vs log<sub>10</sub>HBeAg baseline (WEEK24/WEEK48/WEEK96)
- log<sub>10</sub>HBsAg change from baseline vs log<sub>10</sub> HBeAg change from baseline (WEK24/WEEK48/WEEK96)
- log<sub>10</sub> HbsAg (conventional unit) change from baseline vs ALT (conventional unit) change from baseline (WEEK24/WEEK48/ WEEK96)
- log<sub>10</sub> HBsAg (conventional unit) change from baseline vs HBcrAg (conventional unit) baseline (WEEK24/WEEK48/WEEK96)
- log<sub>10</sub>HbsAg (conventional unit) change from baseline vs HBcrAg (conventional unit) change from baseline (WEEK24/WEEK48/WEEK96)
- log<sub>10</sub>HbsAg (conventional unit) change from baseline vs log<sub>10</sub>HBeAg baseline (WEEK24/WEEK48/WEEK96)
- log<sub>10</sub>HBsAg (conventional unit) change from baseline vs log<sub>10</sub> HBeAg change from baseline (WEEK24/WEEK48/WEEK96)

## 9.4. Background factor of HBsAg Responder/ Non-Responder

To investigate the background factor of HBsAg responder, following summary table on HBsAg responder will be provided

The details of the planned displays are presented in Appendix 12: List of Data Displays.

### Overview of Planned Background factor of HBsAg responder

| [Endpoint / Parameter / Display Type] | Data | Displays Gene | erated |
|---|---|---|---|
| | Table | Figure | Listing |
| Demographic and Baseline Characteristics | | | |
| Demographic Characteristics | Y | | |
| Other Baseline Characteristics | Y | | |
| <b>Medical Conditions and Concomitant Medications</b> | | | |
| Medical Conditions | Y | | |
| Concomitant Medications | Y | | |
| <b>Exposure and Treatment Compliance</b> | | | |
| Treatment compliance | Y | | |
| Exposure to Study Treatment | Y | | |

#### **NOTES:**

• Y = Yes display generated.

## 9.5. Safety Subgroup Analysis

This analysis will be based on the "SP" population, unless otherwise specified. Summary of eGFR,  $\beta$ 2-microglobulin-creatinine ratio, %TRP, Serum Creatine, Serum Phosphorous and Bone density (absolute, %change from baseline) will be provided using subgroup in Section of "5.3.1 Examination of Subgroups".

Summary of eGFR (conventional unit),  $\beta$ 2-microglobulin-creatinine ratio, %TRP, Serum Creatine (conventional unit), Serum Phosphorous (conventional unit) and Bone density (absolute, %change from baseline) will be provided using subgroup (conventional unit) in Section of "5.3.1 Examination of Subgroups".

## 10. REFERENCES

GlaxoSmithKline Document Number 2017N312381\_06: Study Protocol of 205883. A multi-centre, one-arm prospective study to evaluate efficacy and safety of switching from Entecavir (ETV) to Tenofovir Disoproxil Fumarate (TDF) in Japanese chronic hepatitis B HBeAg-positive and HBV-DNA undetectable subjects (5-JUL-2018).

Payne RB, Little AJ, Williams RB, Milner JR: Interpretation of serum calcium levels in patients with abnormal serum proteins. Br Med J 4: 643-646,1973

#### 11. APPENDICES

## 11.1. Appendix 1: Protocol Deviation Management

Details will be referred latest Protocol Deviation Management Plan and data handling will be decided prior to final data base release.

## 11.1.1. Exclusions from Efficacy Evaluable Set

A subject meeting any of the following two criteria will be excluded from the efficacy evaluable set:

Prohibited Medication was taken from start dosing (Beginning of exposure) to week
 48 visit (Date of visit 48 week)

Corresponding prohibited medications are listed as follow. This will be specified as flag 'Y' of DV1 dataset (Excluded from analysis population flag, DVXPPFL) from Data management.

- Interleukin-2 preparations
- Ursodeoxycholic acid preparations
- Herbal medicine with positive effects on hepatic dysfunction
- Antiviral drugs with an inhibitory effect on HBV growth
- Other investigational products
- Interferon preparations
- HB vaccine therapy
- Glucocorticoid preparations (excluding topical preparations such as ointment and cream)
- Immunosuppressants (e.g., azathioprine and cyclophosphamide) or chemotherapeutic agents (e.g., etoposide) (excluding topical preparations such as ointment and cream)
- Treatment compliance from start dosing (Beginning of exposure) to week 48 visit (Date of visit 48 week) was deviated. treatment compliance: <80% or >120%

Corresponding data that prohibited medication was taken will be received by DV1 dataset file from Data management.

Treatment compliance will be calculated from Section 11.6.2 Study Population.

# 11.2. Appendix 2: Schedule of Activities

## 11.2.1. Protocol Defined Schedule of Events

| Procedure | Screening | | | Treatmen | t period | | Discontinuation/Completion |
|---|---|---|---|---|---|---|---|
| | (up to 42<br>days before<br>Day 1) <sup>1</sup> | Day 1 | Week 4<br>(±14) | Week 12, 24, 36 | Week 48<br>(±14) | Week 60, 72, 84<br>(±14) | (Week 96)<br>(±14) <sup>2</sup> |
| | | | | (±14) | | | |
| Informed Consent | X <sup>1</sup> | | | | | | |
| Demography | X | | | | | | |
| Abdominal imaging test <sup>3</sup> | X | (X) | (X) | (X) | (X) | (X) | X |
| Inclusion/Exclusion Criteria <sup>4</sup> | X | | | | | | |
| Pregnancy Test (females of childbearing potential only) <sup>5</sup> | X | X | X | X | X | X | X |
| [HIV and HCV screening] | X | | | | | | |
| 12-lead ECG | X | | | | X | | X |
| Bone densinometry | X <sup>6</sup> | | $(X)^{7,8}$ | $(X)^{7,8}$ | $(X)^{7,8}$ | $(X)^{7,8}$ | X <sup>8</sup> |
| Vital Signs <sup>9</sup> | X | X | X | X | X | X | X |
| Study treatment dispensation | | X | | X | X | X | |
| Confirmation of investigational product compliance | | | X | X | X | X | X |
| AE Assessment | | X | ŧ | | | <b></b> | X |
| SAE Assessment | | X | ŧ | | | | X |
| Concomitant Treatment Review | X | X | ŧ | | | | X |
| Hematology 10 | X | X | X | X | X | X | X |
| Clinical Chemistry 11 | X | X | X | X | X | X | X |
| Urinalysis <sup>12</sup> | X | X | X | X | X | X | X |
| HBV-DNA | X | X | X | X | X | X | X |
| HBeAg/Anti-HBe | X | X | X | X | X | X | X |
| HBsAg/Anti-HBs | X | X | X | X | X | X | X |

| Procedure | Screening | ing Treatment period | | | | Discontinuation/Completion | |
|---|---|---|---|---|---|---|---|
| | (up to 42 | Day 1 | Week 4 | Week 12, 24, | Week 48 | Week 60, 72, 84 | (Week 96) |
| | days before<br>Day 1) <sup>1</sup> | | (±14) | 36<br>(±14) | (±14) | (±14) | (±14) <sup>2</sup> |
| HBcrAg | | X | X | X | X | X | X |
| Resistant Assay 13 | | | (X) | (X) | (X) | (X) | (X) |
| HBV Genotype | X | | | | • | | |

- 1. Perform the screening examinations surely within 42 days before starting the study treatment.
- 2. On completing or discontinuing the study, perform these items within 72 hours after the last dose of the study treatment.
- 3. For diagnosis of cirrhosis, see Appendix 7 in the protocol.
- 4. For subject in whom HBsAg value range is confirmed before screening, enter values at 2 time points (with an interval of at least 3 months, and at least one point within 1 year from screening) into electronic Case Report Form (eCRF).
- 5. Perform the pregnancy test (urine test) for only women of childbearing potential or women with less than two years after the last menstruation. On the day of starting the study treatment, perform the pregnancy test before the first dose of the study treatment.
- 6. If the assessment was performed within 1 year prior to screening, it can be substituted as a score at screening.
- 7. Perform the assessment when the investigator considered necessary from laboratory results.
- 8. Perform bone densimetry with an interval of at least 4 months. If the assessment was performed within 3 months prior to each visit, do not duplicate the procedure.
- 9. Assess height, weight, blood pressure, pulse rate and temperature. Height is collected at screening only.
- 10. Red blood cell count, hemoglobin, hematocrit, white blood cell count (including differential count), platelet count, prothrombin time
- 11. AST, ALT, γ-GTP, ALP, LDH, total bilirubin, direct bilirubin, total protein, serum albumin, serum creatinine, creatinine kinase, amylase, lipase, AFP, antinuclear antibody titer, electrolyte (Na, K, Cl, Ca, P), blood glucose, uric acid, BUN, hyaluronate, lactic acid (however, assess antinuclear antibody titer at screening only, hyaluronate must be assessed at screening but for the visits afterwards assess when necessary), CLcr (calculate from serum creatinine based on Cockcroft-Gault formula described in Section 6.1), eGFR
- 12. Urinary sediment, β2-microglobulin, urine creatinine, urine glucose, urine protein, electrolyte (P)


205883

13. Perform resistance analysis on lamivudine (LAM), adefovir (ADV), ETV and TDF. In a case where a virological breakthrough has been observed (a case where the serum HBV-DNA level has increased from the nadir by at least 1 log IU/mL, or HBV DNA level has increased to ≥2 log IU/mL (100 IU/mL) in a case with nadir <10 IU/mL) perform the resistance analysis. The blood specimen for the resistance analysis must be taken at every visit (excluding the starting date of the study treatment).

## 11.3. Appendix 3: Assessment Windows

## 11.3.1. Definitions of Assessment Windows for Analyses

A) The assessment dates of virology (HBsAg, serum HBV-DNA, HBeAg, HBeAg/Ab, HBsAg/Ab, HBcrAg) and clinical laboratory test for efficacy (i.e. ALT)

| Period | Nominal Day | <b>Lowest Day</b> | Highest Day |
|-----------------|-------------|-------------------|-------------|
| Screening | - | -42 | -1 |
| Baseline (Day1) | 1 | - | 1 |
| Week 4 | 29 | 15 | 43 |
| Week 12 | 85 | 44 | 127 |
| Week 24 | 169 | 128 | 211 |
| Week 36 | 253 | 212 | 295 |
| Week 48 | 337 | 296 | 379 |
| Week 60 | 421 | 380 | 463 |
| Week 72 | 505 | 464 | 547 |
| Week 84 | 589 | 548 | 631 |
| Week 96 | 673 | 632 | 715 |

B) Safety (Laboratory, ECG, Vital Sign and Bone density) data will not be adapted the assessment windows. But 'COMPLETED/WITHDRAWAL' need to be assigned to corresponding visit, by comparing its date with the assessment window. The outsiders, the data being out of any windows will be regarded as 'Unscheduled'

| Period | Nominal Day | Lowest Day | Highest Day |
|-----------------|-------------|------------|-------------|
| Screening | - | -42 | -1 |
| Baseline (Day1) | 1 | - | 1 |
| Week 4 | 29 | 2 | 43 |
| Week 12 | 85 | 44 | 127 |
| Week 24 | 169 | 128 | 211 |

| Period | Nominal Day | <b>Lowest Day</b> | Highest Day |
|---------|-------------|-------------------|-------------|
| Week 36 | 253 | 212 | 295 |
| Week 48 | 337 | 296 | 379 |
| Week 60 | 421 | 380 | 463 |
| Week 72 | 505 | 464 | 547 |
| Week 84 | 589 | 548 | 631 |
| Week 96 | 673 | 632 | 715 |

C) Summary of AE by months will be used below AE occurrence day category (AE for 48 Week report, AE for final CSR).

(AE occurrence day: 48 Week report)

| Months | Days |
|-------------------|-------------------|
| Month 1 | 1 - 29 days |
| Month 2 - 3 | 30 – 85 days |
| Month 4 - 6 | 86 – 169 days |
| Month 7 - 9 | 170 – 253 days |
| Month 10 - 12 | 254 – 337 days |
| Month 13 or later | 338 days or later |

(AE occurrence day: final CSR)

| Months | Days |
|-------------------|-------------------|
| Month 1-12 | 1 - 337 days |
| Month 13- 18 | 338 - 505 days |
| Month 19- 24 | 506 - 673 days |
| Month 25 or later | 674 days or later |

## 11.3.2. Selection of Data in the Event of Multiple Records in a Window

Depending on the statistical method of analysis, single values are required for each analysis window. For example, change from baseline by visit usually requires a single value. When a single value is needed, the following rules will be used based on the type of data that is being analysed.

### 11.3.2.1. Serology, ALT and Laboratory Parameters of Interest

The largest value will be included in the analysis when two or more ALT values occur within the same visit window.
In the event that two or more serology results (HBsAg, HBcrAg, HBeAg, HBsAb, HBeAb) occur within the same visit window, then the pair will remain together and the last pair of results in the window will be chosen.

In the event that multiple observations occur within the same visit window for any other laboratory parameter, the laboratory value (e.g., mg/dL of serum creatinine) that represents the most abnormal value (based on actual value and not on grade) will be used in by-visit summaries for the laboratory parameter. In the event that two values within a window are of equal abnormality (based on actual value and not on grade), the value collected nearest to the nominal date will be used in all summaries.

#### 11.3.2.2. HBV DNA values (log10 IU/mL)

- 1) Select the record closest to the nominal day (e.g. Day 169 for analysis Week 24) for that visit.
- 2) If there are two visits equidistant from the nominal day, take the latest. If there are multiple records on a selected day, take the geometric mean.
- 3) If there are two values on the same day, the second may be a retest because there was a problem with the first test (for example, specimen hemolyzed). In these cases, the later value should be used.

### 11.4. Appendix 4: Study Phases and Treatment States

## 11.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to the assessment date.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date |
| Post-Treatment | Date > Study Treatment Stop Date |

#### 11.4.1.1. Study Phases for Concomitant Medication

| <b>Study Phase</b> | Definition |
|---|---|
| Prior | If medication end date is not missing and is before dosing date. |
| Concomitant | Any medication that is not a prior |

#### **NOTES:**

Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial
dates for concomitant medication. Use the rules in this table if concomitant medication date is
completely missing.

#### 11.4.2. Treatment States for AE data

Adverse events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

| Treatment<br>State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date. |
| | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date |
| Post-Treatment | If AE onset date is after the treatment stop date. |
| | AE Start Date > Study Treatment Stop Date |
| Onset Time | If Treatment Start Date > AE Onset Date: |
| Since 1 <sup>st</sup> Dose | = AE Onset Date - Treatment Start Date |
| (Days) | If Treatment Start Date ≤ AE Onset Date: |
| | = AE Onset Date - Treatment Start Date +1 |
| | Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on eCRF OR value is missing. |

#### **NOTES:**

• If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.

# 11.5. Appendix 5: Data Display Standards & Handling Conventions

### 11.5.1. Reporting Process

| Software | |
|---|---|
| The currently support of the currently su | • The currently supported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | IARP Server N/A |
| HARP Compound | HARP Compound N/A |
| <b>Analysis Datasets</b> | Analysis Datasets |
| Analysis datasets will be created according to Legacy GSK A&R dataset standards | |
| Generation of RTF Files | |
| Non-HARP study. | |

## 11.5.2. Reporting Standards

#### General

• The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### Formats

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.
  - For Insert Endpoint / Parameter the following DP's places will be applied:
  - Summary Statistics:
  - Listings:

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

| Unscheduled Visits | |
|---|---|
| • Unscheduled vi | Unscheduled visits will not be included in summary tables. |
| Unscheduled vi | Unscheduled visits will not be included in figures. |
| All unschedule | All unscheduled visits will be included in listings. |
| <b>Descriptive Summa</b> | Descriptive Summary Statistics |
| Continuous Data | Continuous Data Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data N, n, frequency, % | |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

### 11.6. Appendix 6: Derived and Transformed Data

#### 11.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### **Study Day**

- Calculated as the number of days from administered date:
- Ref Date = Missing

- $\rightarrow$  Study Day = Missing
- Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
- Ref Data  $\geq$  First Dose Date  $\rightarrow$  Study Day = Ref Date (First Dose Date) + 1

### 11.6.2. Study Population

#### **Demographics**

#### Age

- Birth date will be presented in listings as 'YYYY'.
- Reference will be treatment(prescribed) date
- Reference date for age calculation will be from dosing start day (Day 1, Visit 2).
- Reference date for calculation of age at screening will be from Screening visit (Visit 1) date, however this will be from screen failure date for a screen failure subject.
- Analysis age group will be categorized (Years):
  - <=18, 19-64, 65-74, >=75
- Age will be categorized for EudraCT (Years)
  - <=17, 18-64, 65-84, >=85

#### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

#### **Treatment Compliance**

- Compliance (%) will be calculated based on the formula:
  - Compliance (%) = (Prescribed tablet return tablet) / [(Treatment Stop Date Treatment Start Date + 1) x Total daily tablet]
- Subjects who were prescribed but did not report a treatment start date will be categorised as having zero days of exposure.

#### **Treatment Compliance**

• If there are any treatment breaks during the study, exposure data will be adjusted accordingly

e.g. one tablet per 5days, total daily Tablet is 1/5 tablet.

If "As required" in dosing frequency was occurred, previous dosing frequency will be used as calculation.

Image of treatment

| prescribed1 | | Return1 | | Prescribed2 | | Returned2 | |
|-------------|------|---------|------|-------------|------|-----------|------|
| Start1 | End1 | Start2 | End2 | Start3 | End3 | Start4 | End4 |
| 1 x Daily | | Every 3 | days | Every 4 | days | As Requir | red |

• Upper: compliance data, Lower: Exposure data.

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
   Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) +
- Subjects who were prescribed but did not report a treatment start date will be categorised as having zero days of exposure.

### 11.6.3. **Efficacy**

#### HBV- DNA data (log<sub>10</sub> IU/mL)

- HBV DNA data below the LLQ (1.0 log<sub>10</sub>IU/mL) for the assay will be set to the lower limit minus 0.1 (0.9 log<sub>10</sub>IU/mL) for calculation of summary statistics for the actual HBV DNA values and the change from baseline values by study visit. The original values will be provided in the HBV DNA listing.
- Note that if the result will be 'Not detected', that data will be also treated in the same way  $(0.9 \log_{10} IU/mL, 1.0 0.1 \log_{10} IU/mL)$  as the below the LLQ.

#### Virological (HBV-DNA) breakthrough

• In a case where a virological (HBV-DNA) breakthrough has been observed (a case where the serum HBV-DNA level has increased from the nadir by at least 1 log IU/mL, or HBV DNA level has increased to ≥2 log IU/mL (100 IU/mL) in a case with nadir <10 IU/mL) perform the resistance analysis.

#### HBsAg responder/Non-responder

HBsAg reduction potential evaluate ( $log_{10}$  observation –  $log_{10}$  baseline).

HBsAg responder: <=-0.25 log<sub>10</sub> HBsAg Non-responder: >-0.25 log<sub>10</sub>

#### 'Loss' of HBeAg, HBsAg,

'Loss' of HBeAg and HBsAg means antigen is negative.

e.g.

HBsAg Loss %: Numbers of subjects with HBsAg loss / Numbers of subjects with positive HBsAg at baseline

HBeAg Loss %: Numbers of subjects with HBeAg loss / Numbers of subjects with positive HBeAg at baseline

#### Seroconversion of HBsAg and HBeAg

'Seroconversion' of HBsAg and HBeAg means antigen is negative and antibody is positive.

e.g.

HBsAg Seroconversion %: Numbers of subjects with HBsAg/Ab Seroconversion / Numbers of subjects with positive HBsAg and Negative HBsAb at baseline

HBeAg Seroconversion %: Numbers of subjects with HBeAg/Ab Seroconversion / Numbers of subjects with positive HBeAg and Negative HBeAb at baseline

#### HBsAg category

HBsAg is categorised as follow:

<80, 80=< - <800, 800=< - <8000, 8000=< - <80000, >=80000 Unit: KIU/L

#### HBsAg (Conventional unit) category

HBsAg is categorised as follow:

<80, 80=< - <800, 800=< - <8000, 8000=< - <80000, >=80000 Unit: IU/mL

#### HBcrAg category

HBcrAg is categorised as follow:

 $<3.0 \log_{10}, 3.0 = <-<4.0 \log_{10}, 4.0 = <-<5.0 \log_{10}, 5.0 = <-<6.0 \log_{10}, >=6.0 \log_{10}$  Unit: KU/L

#### HBcrAg (conventional unit) category

HBcrAg is categorised as follow:

 $<3.0 \log_{10}, 3.0 = <$  -  $<4.0 \log_{10}, 4.0 = <$  -  $<5.0 \log_{10}, 5.0 = <$  -  $<6.0 \log_{10}, >=6.0 \log_{10}$  Unit: U/mL

### 11.6.4. Safety

#### **Adverse Events**

#### **AEs of Special Interest**

The adverse events of special interest and how they will be identified are outlined below. For more details, Viread (Tenofovir Disoproxil Fumarate) Risk Management Plan for the EU (Version 22, January 2017) or the latest document will be referred (Appendix 10).

- "Renal-AE" Acute renal failure (SMQ), Chronic kidney disease (SMQ), Proteinuria (SMQ) and preferred terms of potentially renal related AEs.
- "Liver AE" Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions (SMQ), Hepatitis, non-infectious (SMQ), Liver related investigations, signs and symptoms (SMQ) and preferred terms of potentially Liver related AEs.
- "Bone Events" Preferred terms of potentially Bone related AEs.

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x' becomes x 0.01
  - o Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - o Example 3: 0 Significant Digits = '< x' becomes x 1

| Laboratory Assessments | |
|---|---|
| Haematology | Platelet Count, RBC Count, Haemoglobin, Hematocrit, Prothrombin time, WBC count with Differential (Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils) |
| Clinical Chemistry | BUN, Creatinine, Glucose, Uric acid, Amylase, Potassium, Sodium, Calcium, Chloride, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline phosphatise, γ-GTP Phosphorus, Total and direct bilirubin, Total Protein, Albumin, LDH, CK (CPK), eGFR, Lipase, AFP, Antinuclear antibody titer [only at the time of screening], Hyaluronic acid [Required at screening and as needed thereafter.], Lactic Acid |
| Routine Urinalysis | Glucose, protein, creatinine, electrolyte (P), urinary sediment, β2-microglobulin |

#### Corrected calcium based on the serum albumin

• Corrected calcium based on the serum albumin will be calculated based on the following Payne formula.

Corrected calcium (mg/dL) = Serum calcium (mg/dL) + [4 - serum albumin (g/dL)], if serum albumin is <4.0 g/dL

#### Consideration of the kidney marker

- $\beta$ 2-microglobulin-creatinine ratio will be calculated based on the following formula. Urinary  $\beta$ 2-microglobulin ( $\mu$ g/g Cre) =100×Urinary  $\beta$ 2-microglobulin ( $\mu$ g/L)/ Urinary creatinine (mg/dL)
- %TRP will be calculated based on the following formula.
   (1 [urinary phosphorus (mg/dL) × serum creatinine (mg/dL)] /. [serum phosphorus (mg/dL) × urinary creatinine (mg/dL)]) × 100

#### Bone density (%)

Bone density (%) = (Bone density observation – Bone density baseline)/ Bone density baseline

#### **Creatinine clearance**

Creatinine clearance (CLcr) formula:

(Body weight [kg]) x (140-age in years) / (72 x serum creatinine [mg/dl]) for man [Note: multiply estimated rate by 0.85 for woman]

#### ECG (12-lead ECG)

ECG findings, ECG values (Heart rate, PR interval, QRS duration, QT interval, and QTc intervals)

#### **Vital Signs**

Pulse rate, Blood pressure (Systolic, Diastolic), Temperature, Weight

#### Gilead Science Institute (GSI) grading laboratory Data

Referred to Gilead Grading Scale for Severity of Laboratory Abnormalities, Laboratory grade frequency will be summarized and listed.

Note that grade tables: We will be referred two tables (Section 11.8.1 LDTA (A Liver Disease Therapeutic Area) GSI grading scale, Section 11.8.2. GSI modified NIAID (National Institute of Allergy and Infectious Disease (US)) Common Toxicity Grading Scale) and displayed. GSI modified NIAID common toxicity grading scale will be applied on the laboratory data to be aligned with foreign clinical studies of Tenofovir.

#### **Abnormality Grades**

Clinical laboratory results will be graded according to criteria specified in the GSI grading score as normal, mild (Grade 1), moderate (Grade 2), severe (Grade 3) or potentially life threatening (Grade 4). Some analytes have criteria for both increased and decreased levels; analysis for each direction (i.e., increased, decreased) will be presented separately. Laboratory abnormalities may be reported as an adverse event, and the clinical grading of an event may be different from the quantitative grading depending on the clinical status and underlying conditions.

#### Gilead Science Institute (GSI) grading laboratory Data

**Treatment-Emergent Abnormalities** 

Treatment-emergent laboratory abnormalities are defined as values that increase at least one grade from baseline at any on-treatment post-baseline visit. If the relevant baseline laboratory data are missing, then the screening laboratory result is used, if this is missing then any graded abnormality is considered treatment emergent.

#### **Treatment-Emergent Marked Abnormalities**

Treatment-emergent marked laboratory abnormalities are defined as values that change from normal at baseline to Grade 3 (severe) or 4 (potentially life threatening) at any post-baseline, on-treatment value, or that change from Grade 1 (mild) at baseline to Grade 4 at any post-baseline. If the relevant baseline laboratory data are missing, then the screening laboratory result is used; if this is missing then any Grade 3 or 4 on-treatment values are considered treatment emergent.

#### Summaries of Laboratory Abnormalities

The following summaries (number and percentage of subjects) of treatment-emergent laboratory abnormalities will be provided:

- (1) Treatment-emergent laboratory abnormalities
- (2) Treatment-emergent Grade 3 or Grade 4 laboratory abnormalities
- (3) Marked laboratory abnormalities
- (4) Incidence of on-treatment exacerbation of hepatitis defined as (1) elevation of ALT > 2 x baseline and > 10 x ULN or (2) abnormal laboratory parameters suggestive of worsening hepatic function (abnormal bilirubin  $\geq 2 \text{mg/dL}$  above baseline, abnormal PT  $\geq$  2 sec above baseline, INR  $\geq$  0.5 over baseline, abnormal albumin  $\geq$  1g/dL decrease from baseline or elevated serum lactate levels > 2 x ULN) along with any ALT elevation (i.e., 1 grade shift or 2 x previous value)

Note that serum lactate is not measured in the study.

- (5) Confirmed (defined as two consecutive visits) increases in serum creatinine of 0.5 mg/dL above baseline
- (6) Confirmed (defined as two consecutive visits) occurrence of phosphorus below 2  $\rm mg/dL$
- (7) Confirmed (defined as two consecutive visits) calculated creatinine clearance < 50 mL/min

# 11.7. Appendix 7: Reporting Standards for Missing Data

# 11.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as described in the Protocol. |
| | Withdrawn subjects were not replaced in the study. |
| | • All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | Withdrawal visits will be slotted as per Appendix 3: |

# 11.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |

# 11.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Partial dates will be displayed as captured in subject listing displays.</li> </ul> |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomita<br>nt<br>Medication<br>s/Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |

| Element | Reporting Detail |
|---------|------------------------------------------------------------|
| | • The recorded partial date will be displayed in listings. |

# 11.7.2.2. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| Withdrawn<br>Subjects | <ul> <li>In analysing the responder analysis, unless otherwise stated, withdrawn subjects reported during the study period will be treated as non-responders.</li> <li>For continuous variables, if subjects will be withdrawn from the study due to adverse events or rescue medication before Week 48/Week 96, data after withdrawal will not be collected, and data analysis will be performed on collected data (i.e. After withdrawal, data will not be collected and data will not be imputed.).</li> </ul> |

# 11.8. Appendix 8: Values of Potential Clinical Importance(PCI)

LDTA GSI grading scale (LDTA GSI grade), GSI modified NIAID Common Toxicity Grading Scale (GSI NIAID grade) will be treated as PCI.

# 11.8.1. LDTA GSI grading scale (LDTA GSI grade)

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hemoglobin | 10.0 to 10.9<br>g/dL | 9.0 to < 10.0 g/dL | 7.0 to < 9.0 g/dL | < 7.0 g/dL |
| [Hemoglobin] | 100 to 109 g/L | 90 to < 100 g/L | 70 to < 90 g/L | < 70 g/L |
| | OR | OR | OR | |
| | Any decrease from Baseline | Any decrease from Baseline | Any decrease from Baseline | |
| | 2.5 to < 3.5 g/dL | 3.5 to < 4.5 g/dL | $\geq 4.5 \text{ g/dL}$ | |
| | 25 to < 35 g/L | 35 to < 45 g/L | ≥ 45 g/L | |
| Absolute<br>Neutrophil Count | 1000 to<br>1300/mm <sup>3</sup> | 750 to < 1000/mm <sup>3</sup> | 500 to < 750/mm <sup>3</sup> | < 500/mm <sup>3</sup> |
| (ANC) | 1.00 to 1.30<br>GI/L | 0.75 to < 1.00<br>GI/L | 0.50 to < 0.75<br>GI/L | < 0.50 GI/L |
| [-] | | | | |
| Absolute<br>Lymphocyte | 600 to 650/mm <sup>3</sup> | $500 \text{ to} < 600/\text{mm}^3$ | 350 to < 500/mm <sup>3</sup> | < 350/mm <sup>3</sup> |
| Count [-] | 0.60 to 0.65<br>GI/L | 0.50 to < 0.60<br>GI/L | 0.35 to < 0.50<br>GI/L | < 0.35 GI/L |
| L J | | | OI/L | |
| Platelets | 100,000 to < 125,000/mm <sup>3</sup> | 50,000 to < 100,000/mm <sup>3</sup> | 25,000 to < 50,000/mm <sup>3</sup> | < 25,000/mm <sup>3</sup> |
| [Platelet count] | 100 to < 125<br>GI/L | 50 to < 100 GI/L | 25 to < 50 GI/L | < 25 GI/L |
| WBCs | 2000/mm <sup>3</sup> to 2500/mm <sup>3</sup> | 1,500 to < 2,000/mm <sup>3</sup> | 1000 to < 1,500/mm <sup>3</sup> | < 1000/mm <sup>3</sup> |
| [WBC] | 2.00 GI/L to<br>2.50 GI/L | 1.50 to < 2.00<br>GI/L | 1.00 to < 1.50<br>GI/L | < 1.00 GI/L |

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Prothrombin Time (PT) [ Prothrombin Time] | > 1.00 to 1.25 × ULN | > 1.25 to 1.50 ×<br>ULN | > 1.50 to 3.00 × ULN | > 3.00 × ULN |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyponatremia<br>[Sodium] | 130 to 135<br>mEq/L | 125 to < 130<br>mEq/L | 121 to < 125<br>mEq/L | < 121 mEq/L |
| | 130 to 135<br>mmol/L | 125 to < 130<br>mmol/L | 121 to < 125<br>mmol/L | < 121 mmol/L |
| Hypernatremia [Sodium] | 146 to 150<br>mEq/L | > 150 to 154<br>mEq/L | > 154 to 159<br>mEq/L | > 159 mEq/L |
| | 146 to 150<br>mmol/L | > 150 to 154<br>mmol/L | > 154 to 159<br>mmol/L | > 159 mmol/L |
| Hypokalemia<br>[Potassium] | 3.0 to 3.4 mEq/L | 2.5 to < 3.0<br>mEq/L | 2.0 to < 2.5<br>mEq/L | < 2.0 mEq/L |
| | 3.0 to 3.4<br>mmol/L | 2.5 to < 3.0<br>mmol/L | 2.0 to < 2.5<br>mmol/L | < 2.0 mmol/L |
| Hyperkalemia<br>[Potassium] | 5.6 to 6.0 mEq/L | > 6.0 to 6.5<br>mEq/L | > 6.5 to 7.0<br>mEq/L | > 7.0 mEq/L |
| | 5.6 to 6.0<br>mmol/L | > 6.0 to 6.5<br>mmol/L | > 6.5 to 7.0<br>mmol/L | > 7.0 mmol/L |
| Hypoglycemia<br>[Glucose] | 55 to 64 mg/dL<br>3.03 to 3.58<br>mmol/L | 40 to < 55 mg/dL<br>2.20 to < 3.03<br>mmol/L | 30 to < 40 mg/dL<br>1.64 to < 2.20<br>mmol/L | < 30 mg/dL<br>< 1.64 mmol/L |
| Hyperglycemia,<br>Nonfasting | 116 to 160<br>mg/dL | > 160 to 250<br>mg/dL | > 250 to 500<br>mg/dL | > 500 mg/dL |
| [Glucose] | 6.42 to 8.91<br>mmol/L | > 8.91 to 13.90<br>mmol/L | > 13.90 to 27.79<br>mmol/L | > 27.79<br>mmol/L |
| Hypocalcemia [Calcium] (corrected for albumin) | 7.8 to 8.4 mg/dL | 7.0 to < 7.8<br>mg/dL | 6.1 to < 7.0 mg/dL | < 6.1 mg/dL |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hypercalcemia [Calcium] (corrected for albumin) | 10.6 to 11.5<br>mg/dL | > 11.5 to 12.5<br>mg/dL | > 12.5 to 13.5 mg/dL | > 13.5 mg/dL |
| Hypophosphatemia [Phosphorous?] | NA | 2.0 to < 2.5 mg/dL | 1.0 to < 2.0 mg/dL | < 1.0 mg/dL |
| | | 0.63 to < 0.80<br>mmol/L | 0.31 to < 0.63<br>mmol/L | < 0.31 mmol/L |
| Hyperbilirubinemia [Total bilirubin?] | > 1.0 to 1.5 ×<br>ULN | > 1.5 to 2.5 ×<br>ULN | > 2.5 to 5.0 ×<br>ULN | > 5.0 × ULN |
| Blood Urea<br>Nitrogen<br>[BUN] | 1.25 to 2.50 ×<br>ULN | > 2.50 to 5.00 ×<br>ULN | > 5.00 to 10.00 ×<br>ULN | > 10.00 × ULN |
| Creatinine [Creatinine] | > 1.50 to 2.00<br>mg/dL<br>> 133 to 177<br>µmol/L | > 2.00 to 3.00<br>mg/dL<br>> 177 to 265<br>µmol/L | > 3.00 to 6.00<br>mg/dL<br>> 265 to 530<br>µmol/L | $> 6.00$ mg/dL $> 530$ $\mu$ mol/L |
| Creatine Kinase [CK] | 3.0 to < 6.0 ×<br>ULN | 6.0 to < 10.0 ×<br>ULN | 10.0 to < 20.0 ×<br>ULN | ≥ 20.0 × ULN |

| ENZYMES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| AST (SGOT) [AST] | 1.25 to 2.50 ×<br>ULN | > 2.50 to 5.00 ×<br>ULN | > 5.00 to 10.00 ×<br>ULN | > 10.00 × ULN |
| ALT (SGPT) [ALT] | 1.25 to 2.50 ×<br>ULN | > 2.50 to 5.00 ×<br>ULN | > 5.00 to 10.00 ×<br>ULN | > 10.00 × ULN |
| Alkaline<br>Phosphatase<br>[ALP] | 1.25 to 2.50 ×<br>ULN | > 2.50 to 5.00 ×<br>ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |

| ENZYMES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Total Amylase [Amylase] | > 1.0 to 1.5 ×<br>ULN | > 1.5 to 2.0 ×<br>ULN | > 2.0 to 5.0 ×<br>ULN | > 5.0 × ULN |
| Albumin [Albumin] | 3.0 g/dL to <<br>LLN<br>30 g/L to < LLN | 2.0 to < 3.0 g/dL<br>20 to < 30 g/L | < 2.0 g/dL<br>< 20 g/L | NA |

ULN = Upper Limit of Normal; LLN = Lower Limit of Normal

Although Section 11.8.1 mentioned unit for electrolyte Ca is "mg/dL", these values were converted values based on "mmol/L" unit that is used as one of GSK SI units. For laboratory grading, following grades in the table has been applied.

| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Hypocalcemia [Calcium] | 1.94 to 2.10<br>mmol/L | 1.74 to 1.94<br>mmol/L | 1.51 to 1.74<br>mmol/L | 1.51 mmol/L |
| (corrected for albumin) | | | | |
| Hypercalcemia [Calcium] (corrected for albumin) | 2.64 to 2.88<br>mmol/L | 2.88 to 3.13<br>mmol/L | 3.13 to 3.38<br>mmol/L | 3.38 mmol/L |

# **11.8.2.** GSI modified NIAID Common Toxicity Grading Scale (GSI NIAID grade)

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hemoglobin | 8.0 – 9.4 g/dL<br>80 – 94 g/L | 7.0 - < 8.0 g/dL<br>70 - < 80 g/L | 6.5-<7.0 g/dL<br>65-<70 g/L | < 6.5 g/dL<br>< 65 g/L |
| [Hemoglobin] | , , , , g, <u>z</u> | 70 00 8/2 | 70 82 | 30 8/2 |
| Platelets | 75,000 – | 50,000 - < | 25,000 - < | < 25,000/mm3 |
| | 100,000/mm3 | 75,000/mm3 | 50,000/mm3 | < 25.0 GI/L |
| [Platelet count] | 75.0 - 100.0 | 50.0 - < 75.0 GI/L | 25.0 - < 50.0 | |
| | GI/L | | GI/L | |

<sup>[-]:</sup> Not measured

LDTA: Liver Disease Therapeutic Area (Toxicity Grading Scale)

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| WBCs | 3000/mm3- <<br>LLN | 2000 – <<br>3000/mm3 | 1000 – <<br>2000/mm3 | < 1000/ mm3<br>< 1.0 GI/L |
| [WBC] | 3.0 GI/L - <<br>LLN | 2.0 - < 3.0 GI/L | 1.0 - < 2.0 GI/L | |
| Prothrombin Time (PT) | > 1.00 – 1.25 ×<br>ULN | > 1.25 – 1.50 ×<br>ULN | > 1.50 – 3.00 ×<br>ULN | > 3.00 × ULN |
| [Prothrombin<br>Time] | | | | |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyponatremia | 130 mEq/L - < | 123-< 130 | 116 – < 123 | < 116 mEq/L |
| | LLN | mEq/L | mEq/L | < 116 mmol/L |
| [Sodium] | 130 mmol/L – < | 123-< 130 | 116 - < 123 | |
| | LLN | mmol/L | mmol/L | |
| Hypernatremia | > ULN – 150 | > 150 – 157 | > 157 – 165 | > 165 mEq/L |
| | mEq/L | mEq/L | mEq/L | > 165 mmol/L |
| [Sodium] | > ULN – 150 | > 150 – 157 | > 157 – 165 | |
| | mmol/L | mmol/L | mmol/L | |
| Hypokalemia | 3.0 mEq/L - < | 2.5 - < 3.0 mEq/L | 2.0 - < 2.5 | < 2.0 mEq/L |
| | LLN | 2.5 - < 3.0 | mEq/L | < 2.0 mmol/L |
| [Potassium] | 3.0 mmol/L - < | mmol/L | 2.0 - < 2.5 | |
| | LLN | | mmol/L | |
| Hyperkalemia | 5.6 - 6.0 mEq/L | > 6.0 - 6.5 mEq/L | > 6.5 – 7.0 | > 7.0 mEq/L |
| FD : 1 | 5.6 - 6.0 | > 6.0 - 6.5 | mEq/L | > 7.0 mmol/L |
| [Potassium] | mmol/L | mmol/L | > 6.5 - 7.0 | |
| ** 1 | 7.7 CA /17 | 40 55 /17 | mmol/L | 20 / 17 |
| Hypoglycemia | 55 - 64 mg/dL | 40 - < 55 mg/dL | 30 - < 40 mg/dL | < 30 mg/dL |
| FC1 1 | 3.03 - 3.57 | 2.20 - < 3.03 | 1.64 - < 2.20 | < 1.64 mmol/L |
| [Glucose] | mmol/L | mmol/L | mmol/L | |
| Hyperglycemia | > ULN – 160 | > 160 - 250 | > 250 - 500 | > 500 mg/dL |
| (nonfasting and | mg/dL | mg/dL | mg/dL | > 27.77 |
| no prior diabetes) | > ULN - 8.90 | > 8.90 – 13.90 | > 13.90 – 27.77 | mmol/L |
| | mmol/L | mmol/L | mmol/L | |
| [Glucose] | | | | |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hypocalcemia<br>(corrected for<br>albumin)<br>[Calcium] | 7.8 mg/dL - <<br>LLN<br>1.94 mmol/L - <<br>LLN | 7.0 - < 7.8 mg/dL<br>1.74 - < 1.94<br>mmol/L | 6.1 - < 7.0<br>mg/dL<br>1.52 - < 1.74<br>mmol/L | < 6.1 mg/dL<br>< 1.52 mmol/L |
| Hypercalcemia<br>(corrected for<br>albumin)<br>[Calcium] | > ULN - 11.5<br>mg/dL<br>> ULN - 2.88<br>mmol/L | > 11.5 – 12.5<br>mg/dL<br>> 2.88 – 3.13<br>mmol/L | > 12.5 – 13.5<br>mg/dL<br>> 3.13 – 3.38<br>mmol/L | > 13.5 mg/dL<br>> 3.38 mmol/L |
| Hypophosphatemia [Phosphorous] | 2.0 mg/dL - <<br>LLN<br>0.63 mmol/L - <<br>LLN | 1.5 - < 2.0 mg/dL<br>0.47 - < 0.63<br>mmol/L | 1.0 - < 1.5<br>mg/dL<br>0.31 - < 0.47<br>mmol/L | < 1.0 mg/dL<br>< 0.31 mmol/L |
| Hyperbilirubinemia [Total Bilirubin] | > 1.0 – 1.5 ×<br>ULN | > 1.5 – 2.5 × ULN | > 2.5 – 5.0 ×<br>ULN | > 5.0 × ULN |
| Blood Urea<br>Nitrogen | 1.25 – 2.50 ×<br>ULN | > 2.50 – 5.00 ×<br>ULN | > 5.00 – 10.00 ×<br>ULN | > 10.00 × ULN |
| [Urea/BUN] | | | | |
| Hyperuricemia [Uric acid] | > ULN - 10.0<br>mg/dL<br>> ULN - 0.59<br>mmol/L | > 10.0 - 12.0<br>mg/dL<br>> 0.59 - 0.71<br>mmol/L | > 12.0 - 15.0<br>mg/dL<br>> 0.71 - 0.89<br>mmol/L | > 15.0 mg/dL<br>> 0.89 mmol/L |
| Hypouricemia<br>[Uric acid] | 1.5 mg/dL - <<br>LLN<br>0.09 mmol/L - <<br>LLN | 1.0 - <1.5 mg/dL<br>0.06 - < 0.09<br>mmol/L | 0.5 - < 1.0<br>mg/dL<br>0.03 - < 0.06<br>mmol/L | < 0.5 mg/dL<br>< 0.03 mmol/L |
| Creatinine [Creatinine] | M: >1.5 - 2.0<br>mg/dL<br>F: >1.3 - 1.8<br>mg/dL<br>M: >137 - 181<br>micromol/L<br>F: >119 - 163<br>micromol/L | M: > 2.0 - 3.0<br>mg/dL<br>F: > 1.8 - 2.8<br>mg/dL<br>M: > 181 - 269<br>micromol/L<br>F: > 163 - 252<br>micromol/L | M: > 3.0 - 6.0<br>mg/dL<br>F: > 2.8 - 5.8<br>mg/dL<br>M: > 269 - 535<br>micromol/L<br>F: > 252 - 517<br>micromol/L | M: > 6.0<br>mg/dL<br>F: > 5.8 mg/dL<br>M: > 535<br>micromol/L<br>F: > 517<br>micromol/L |
| Creatine Kinase [Creatine Kinase/CK(CPK)] | 3.0 - < 6.0 ×<br>ULN | 6.0 – < 10.0 ×<br>ULN | 10.0 - < 20.0 ×<br>ULN | ≥ 20.0 × ULN |

| ENZYMES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| AST (SGOT) [AST] | 1.25 – 2.50 ×<br>ULN | > 2.50 – 5.00 ×<br>ULN | > 5.00 – 10.00 ×<br>ULN | > 10.00 × ULN |
| ALT (SGPT) [ALT] | 1.25 – 2.50 ×<br>ULN | > 2.50 – 5.00 ×<br>ULN | > 5.00 – 10.00 ×<br>ULN | > 10.00 × ULN |
| GGT<br>[GGT] | 1.25 – 2.50 ×<br>ULN | > 2.50 – 5.00 ×<br>ULN | > 5.00 – 10.00 ×<br>ULN | > 10.00 × ULN |
| Alkaline<br>Phosphatase<br>[ALP] | 1.25 – 2.50 ×<br>ULN | > 2.50 – 5.00 ×<br>ULN | > 5.00 – 10.00 ×<br>ULN | > 10.00 × ULN |
| Total Amylase [Amylase] | > 1.0 – 1.5 ×<br>ULN | > 1.5 – 2.0 × ULN | > 2.0 – 5.0 ×<br>ULN | > 5.0 × ULN |
| Lipase<br>[Lipase] | > 1.0 – 1.5 ×<br>ULN | > 1.5 – 2.0 × ULN | > 2.0 – 5.0 ×<br>ULN | > 5.0 × ULN |
| Albumin [Albumin] | 3.0 g/dL - <<br>LLN<br>30 g/L - < LLN | 2.0 - < 3.0 g/dL<br>20 - < 30 g/L | < 2.0 g/dL<br>< 20 g/L | _ |

ULN = Upper Limit of Normal; LLN = Lower Limit of Normal [-]: not measured in the study

NIAID: National Institute of Allergy and Infectious Disease (US)

# 11.9. Appendix 9: PEGINTERFERON GSKDrug codes

| Term Name | Code |
|-----------------------------------|----------|
| PEGINTERFERON ALFA-2B + RIBAVIRIN | 53239301 |
| PEGINTERFERON NOS | 53332901 |
| PEGINTERFERON ALFA-2A | 51080801 |
| PEGINTERFERON ALFA | 59758801 |
| PEGINTERFERON ALFA-2B | 51090301 |
| PEGINTERFERON BETA 1A | 59122901 |
| PEGINTERFERON ALFA-2A + RIBAVIRIN | 53239401 |
| PEGINTERFERON ALFA | 59758801 |
| PEGINTERFERON ALFA-2A | 51080801 |
| PEGINTERFERON ALFA-2A + RIBAVIRIN | 53239401 |
| PEGINTERFERON ALFA-2B | 51090301 |
| PEGINTERFERON ALFA-2B + RIBAVIRIN | 53239301 |
| PEGINTERFERON BETA 1A | 59122901 |
| PEGINTERFERON LAMBDA-1A | 59611101 |
| PEGINTERFERON NOS | 53332901 |
| ROPEGINTERFERON ALFA-2B | 59745201 |

# 11.10. Appendix 10: Viread (Tenofovir Disoproxil Fumarate) Risk Management Plan for the EU (Version 22) January 2017

MedDRA terms (Version 17.0)

#### Renal toxicity

MedDRA terms (Version 19.1)

SMOs: Acute renal failure, Chronic kidney disease, Proteinuria PTs: Alpha 1 microglobulin urine increased, Computerised tomogram kidney abnormal, Perinephritis, Beta 2 microglobulin abnormal, Beta 2 microglobulin decreased, Beta 2 microglobulin urine abnormal, Blood magnesium abnormal, Blood magnesium decreased, Blood phosphorus decreased, Blood potassium decreased, Blood uric acid abnormal, Blood uric acid decreased, Cystatin C abnormal, Cystatin C increased, Fanconi syndrome, Fanconi syndrome acquired, Glucose urine present, Glycosuria, Henoch-Schonlein purpura nephritis, Hepatorenal syndrome, Renal transplant failure, Hypercalciuria, Hyperchloraemia, Hyperkaliuria, Hypermagnesuria, Hyperphosphaturia, Hyperuricosuria, Hypokalaemia, Hypophosphataemia, Hypouricaemia, Inulin renal clearance abnormal, Nephritis allergic, Nephrogenic diabetes insipidus, Nocturia, Pollakiuria, Polydipsia, Polyuria, Renal disorder, Renal injury, Renal tubular acidosis. Tubulointerstitial nephritis and uveitis syndrome. Urine calcium increased, Urine calcium/creatinine ratio increased, Urine electrolytes abnormal, Urine electrolytes increased, Urine magnesium increased, Urine output increased, Urine phosphorus abnormal, Urine phosphorus increased, Urine potassium abnormal, Urine potassium increased, Urine sodium abnormal, Urine sodium increased, Urine uric acid abnormal, Urine uric acid increased

#### Bone Events due to Proximal Renal Tubulopathy/Loss of Bone Mineral Density (BMD)

MedDRA terms (Version 19.1) HLGT: Fractures

HLT: Fracture treatments (excl skull and spine)

PTs: Bedridden, Blood 25-hydroxycholecalciferol decreased, Blood alkaline phosphatase increased, Bone atrophy, Bone decalcification, Bone densitometry, Bone density abnormal, Bone density decreased, Bone development abnormal, Bone disorder, Bone erosion, Bone formation test abnormal, Bone formation decreased, Bone fragmentation, Bone lesion, Bone loss, Bone metabolism disorder, Bone marrow oedema, Bone marrow oedema syndrome, Bone pain, Bone resorption test abnormal, Bone scan abnormal, Bone swelling, Cementoplasty, Chronic kidney disease – mineral and bone disorder, Coccydynia, C-telopeptide increased, Deoxypyridinoline urine increased, Elevation skull fracture, Fracture pain, High turnover osteopathy, Hip arthroplasty, Hungry bone syndrome, Hypophosphataemic rickets, Immobile, Immobilisation prolonged, Kyphoscoliosis, Kyphosis, Locomotive syndrome, N-telopeptide urine abnormal, N-telopeptide urine increased, Nuclear magnetic resonance imaging spinal abnormal, Osteocalcin increased, Osteodystrophy, Osteolysis, Osteomalacia, Osteopenia, Osteoporosis, Osteoporosis circumscripta

cranii, Osteoporosis menopausal, Osteoporosis prophylaxis, Osteosynthesis, Post-traumatic osteoporosis, Pubic pain, Pyridinoline urine increased, Rachitic syndrome, Renal rickets, Resorption bone increased, Rickets, Senile osteoporosis, Skeletal injury, Skeletal survey abnormal, Spinal deformity, Spinal flattening, Spinal fusion fracture, Spinal X-ray abnormal, Surgical fixation of rib fracture, Tartrate-resistant acid phosphate decreased, Vertebral body replacement, Vertebral lesion, Vertebral wedging, Vertebroplasty, Vitamin D abnormal, Vitamin D decreased, Vitamin D deficiency, Walking aid user, Walking disability, Wheelchair user, X-ray limb abnormal, X-ray of pelvis and hip abnormal, Pain in jaw

#### Post-Treatment Hepatic Flares in HBV Monoinfected and HIV-1/HBV Coinfected Patients

MedDRA terms (Version 19.1) <u>SMQs</u>: Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions; Hepatitis, non-infectious; Liver related investigations, signs and symptoms

PTs: Acute hepatitis B, Asymptomatic viral hepatitis, Chronic disease, Chronic hepatitis B, Concomitant disease aggravated, Concomitant disease progression, Condition aggravated, Disease progression, Disease recurrence, HBV-DNA polymerase increased, HBV-DNA polymerase increased, Hepatitis B, Hepatitis B antibody abnormal, Hepatitis B antibody positive, Hepatitis B core antibody positive, Hepatitis B core antibody positive, Hepatitis B core antipody positive, Hepatitis B e antipody positive, Hepatitis B e antigen positive, Hepatitis B surface antigen positive, Hepatitis B virus test positive, Hepatitis infectious, Hepatitis viral, Hepatitis viral test positive, Hepatobiliary infection, Jaundice, Rebound effect, Viral load increased, Viral titre increased, Withdrawal hepatitis

# 11.11. Appendix 11: Abbreviations & Trade Marks

# 11.11.1. Abbreviations

| Abbreviation | Description |
|--------------|-----------------------------------------------------------|
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| CI | Confidence Interval |
| CLcr | Creatinine Clearance |
| CSR | Clinical Study Report |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| GSI | Gilead Science Institute |
| GSK | GlaxoSmithKline |
| HARP | Harmonisation for Analysis and Reporting Program |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| IP | Investigational Product |
| LDTA | Liver Disease Therapeutic Area (Toxicity Grading Scale) |
| NIAID | National Institute of Allergy and Infectious Disease (US) |
| PCI | Potential Clinical Importance |
| PDMP | Protocol Deviation Management Plan |
| QC | Quality Control |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SOP | Standard Operation Procedure |
| TFL | Tables, Figures & Listings |

# 11.11.2. Trademarks

| Trademarks of the GlaxoSmithKlin<br>Group of Companies | e |
|--------------------------------------------------------|---|
| None | |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
| Viread |

### 11.12. Appendix 12: List of Data Displays

## 11.12.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.1 to 1.23 | - |
| Efficacy | 2.1 to 2.61 | 2.1 to 2.15 |
| Safety | 3.1 to 3.40 | 3.1 to 3.10 |
| Exploratory | 4.1 to 4.42 | 4.1 to 4.48 |
| Section | Listings | |
| ICH Listings | 1 to 72 | |

### 11.12.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 13: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |

#### **NOTES:**

• Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 11.12.3. Deliverables

| Delivery Priority <sup>1</sup> | Description |
|--------------------------------|-------------------------------------------|
| SAC [1] | 48W Statistical Analysis Complete |
| SAC [2] | 96W (Final) Statistical Analysis Complete |

#### **NOTES:**

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 11.12.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | Safety | ES1 | Summary of Subject Disposition | Completed or withdrawn and the reason for withdrawal. | SAC [1,2] |
| 1.2. | Enrolled | ES6 | Summary of Screening Status and Reasons for Screen Failure | The number (%) of Prescribed or screening failure subjects as the screening status, and the reason for screening failure. | SAC [1,2] |
| Protoc | ol Deviation | | | | |
| 1.3. | Safety | IE1 | Summary of Inclusion/Exclusion Criteria Deviations | | SAC [1,2] |
| 1.4. | Safety | DV1 | Summary of Important Protocol Deviations (48W/96W) | | SAC [1,2] |
| Popula | tion Analysed | l | | | |
| 1.5. | Enrolled | SP1 | Summary of Study Populations (48W/96W) | | SAC [1,2] |
| Demog | graphic and B | aseline Charact | eristics | | |
| 1.6. | Safety | DM1 | Summary of Demographic Characteristics (SP) | Age category:<=18, 19-64, 65-74, >=75 | SAC [1,2] |
| 1.7. | FAS | DM1 | Summary of Demographic Characteristics (FAS) | Age category:<=18, 19-64, 65-74, >=75 | SAC [1,2] |
| 1.8. | EES | DM1 | Summary of Demographic Characteristics (EES,48W) | Age category:<=18, 19-64, 65-74, >=75 | SAC [1] |
| 1.9. | Screening<br>Failure | DM1 | Summary of Demographic Characteristics for Screening Failure | Age category:<=18, 19-64, 65-74, >=75 | SAC [1] |
| 1.10. | Enrolled | DM11 | Summary of Age Ranges | <=17, 18-64, 65-84, >=85 | SAC [1,2] |

| Study | Population Ta | ables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.11. | Safety | DM5 | Summary of Race and Racial Combinations (SP) | | SAC [1,2] |
| 1.12. | FAS | DM5 | Summary of Race and Racial Combinations (FAS) | | SAC [1,2] |
| 1.13. | EES | DM5 | Summary of Race and Racial Combinations (EES, 48W) | | SAC [1] |
| 1.14. | Safety | Study specific | Summary of Other Baseline Characteristics (SP) | Include eGFR Subgroup category<br>Genotype categories (A, B, C, D) | SAC [1,2] |
| 1.15. | FAS | Study specific | Summary of Other Baseline Characteristics (FAS) | Include Subgroup category Genotype categories (A, B, C, D) | SAC [1,2] |
| 1.16. | EES | Study specific | Summary of Other Baseline Characteristics (EES,48W) | Include Subgroup category Genotype categories (A, B, C, D) | SAC [1] |
| Prior a | and Concomit | ant Medications | | | 1 |
| 1.17. | Safety | MH4 | Summary of Prior Medical Conditions | | SAC [1,2] |
| 1.18. | Safety | CM1 | Summary of Prior Hepatitis Medications | | SAC [1,2] |
| 1.19. | Safety | CM1 | Summary of Concomitant Medications | | SAC [1,2] |
| Expos | ure and Treat | ment Complian | ce | | |
| 1.20. | FAS | Study specific | Summary of Treatment compliance (FAS) | Note: calculation formula Sum of [(IPCOMPLY.DISPNUM - IPCOMPLY.RETRNNUM)] / sum of [(EXPOSURE.EXENDT - EXPOSURE.EXSTDT + 1) × 1] "Sum of" is cumulative visit | SAC [1,2] |
| 1.21. | EES | Study specific | Summary of Treatment compliance (EES,48W) | | SAC [1] |

| Study 1 | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.22. | Safety | EX1 | Duration of Exposure to Study Drug (SP) | | SAC [1,2] |
| Subgro | oup | | | | |
| 1.23. | FAS | Study specific | Summary of Other Baseline Characteristics by subgroup (FAS) | Protocol defined liver cirrhosis (Yes, No), Genotype (A, B, C, D), HBsAg subgroup category (<800 KIU/L, >=800 KIU/L), AGE category (<40, 40-49, 50-59, 60-), Former Peg-INF (Yes, No) HBsAg subgroup category with conventional unit) (<800 IU/mL, >=800 IU/mL) | SAC [1,2] |

# 11.12.5. Efficacy Tables

| Effica | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prima | ry Endpoint: | HBsAg | | | |
| 2.1. | FAS | Study specific | Proportion of subjects with HBsAg achieving 0.25 Log10 HBsAg reduction from the baseline (HBsAg responder) (FAS,48W, Missing at worse) | Proportion with 95% CI | SAC [1] |
| 2.2. | EES | Study specific | Proportion of subjects with HBsAg achieving 0.25 Log10 HBsAg reduction from the baseline (HBsAg responder) (EES,48W, Missing at worse) | Proportion with 95% CI | SAC [1] |
| 2.3. | FAS | Study specific | Summary of log10 HBsAg (Baseline, FAS) | | SAC [1] |
| 2.4. | EES | Study specific | Summary of log10 HBsAg (Baseline, EES) | | SAC [1] |
| 2.5. | FAS | Study specific | Proportion of subjects with HBsAg achieving 0.25 Log10 HBsAg reduction from the baseline by Subgroup (FAS, 48W/96W, Missing at worse) | Protocol defined Liver cirrhosis (Yes, No), Genotype (A, B, C, D), HBsAg subgroup category (<800 KIU/L, >=800 KIU/L), AGE category (<40, 40-49, 50-59, 60-), Former Peg-INF (Yes, No), HBsAg subgroup category (Conventional unit) (<800 IU/mL, >=800 IU/mL) Proportion with 95% CI | SAC [1,2] |
| 2.6. | EES | Study specific | Proportion of subjects with HBsAg achieving 0.25 Log10 HBsAg reduction from the baseline by Subgroup (EES, 48W, Missing at worse) | Protocol defined liver cirrhosis (Yes, No), Genotype (A, B, C, D), HBsAg subgroup category (<800 KIU/L, >=800 KIU/L), AGE category (<40, 40-49, 50-59, 60-), Former Peg-INF (Yes, No), HBsAg subgroup category (Conventional unit) (<800 IU/mL, >=800 IU/mL) Proportion with 95% CI | SAC [1] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Second | lary Endpoint | t: HBsAg | | | • |
| 2.7. | FAS | Study specific | Proportion of subjects with HBsAg achieving 0.25 Log10 HBsAg reduction from the baseline (HBsAg responder) by study visit up to WEEK 48/WEEK 96 (FAS, Missing at worse) | Proportion with 95% CI | SAC [1,2] |
| 2.8. | FAS | Study specific | Summary of log10 HBsAg by study visit up to WEEK 48/WEEK 96 (FAS) | Change from baseline is included. | SAC [1,2] |
| 2.9. | EES | Study specific | Summary of log10 HBsAg by study visit up to WEEK 48 (EES) | Change from baseline is included. | SAC [1] |
| 2.10. | FAS | Study specific | Summary of HBsAg by study visit up to WEEK 48/WEEK 96 (FAS) | Change from baseline is included. | SAC [1,2] |
| 2.11. | EES | Study specific | Summary of HBsAg by study visit up to WEEK 48 (EES) | Change from baseline is included. | SAC [1] |
| 2.12. | FAS | Study specific | Frequency of HBsAg category by study visit up to WEEK 48/WEEK 96 (FAS) | HBsAg category: <80, 80<= -<br><800, 800<= - <8000, 8000<= -<br><80000, >=80000 Unit: KIU/L | SAC [1,2] |
| 2.13. | EES | Study specific | Frequency of HBsAg category by study visit up to WEEK 48 (EES) | HBsAg category: <80, 80<= -<br><800, 800<= - <8000, 8000<= -<br><80000, >=80000 Unit: KIU/L | SAC [1] |
| 2.14. | FAS | Study specific | Summary of log10 HBsAg (Conventional unit) by study visit up to WEEK 48/WEEK 96 (FAS) | Change from baseline is included. | SAC [1,2] |
| 2.15. | FAS | Study specific | Summary of HBsAg (Conventional unit) by study visit up to WEEK 48/WEEK 96 (FAS) | Change from baseline is included. | SAC [1,2] |
| 2.16. | FAS | Study specific | Frequency of HBsAg category (Conventional unit) by study visit up to WEEK 48/WEEK 96 (FAS) | HBsAg category: <80, 80<= -<br><800, 800<= - <8000, 8000<= -<br><80000, >=80000 Unit: IU/mL | SAC [1,2] |
| Seroco | nversion | | | | |
| 2.17. | FAS | Study specific | Proportion of subjects with HBsAg Loss by Study Visit up to WEEK 48/WEEK 96 (FAS) | % Numbers of subjects with<br>HBsAg loss/Numbers of subjects<br>with positive HBsAg at baseline | SAC [1,2] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.18. | EES | Study specific | Proportion of subjects with HBsAg Loss by Study Visit up to WEEK 48 (EES) | % Numbers of subjects with HBsAg loss/Numbers of subjects with positive HBsAg at baseline | SAC [1] |
| 2.19. | FAS | Study specific | Proportion of subjects with HBsAg/Ab Seroconversion by Study Visit up to WEEK 48/WEEK 96 (FAS) | % Numbers of subjects with HBsAg/Ab Seroconversion/Numbers of subjects with positive HBsAg and Negative HBsAb at baseline | SAC [1,2] |
| 2.20. | EES | Study specific | Proportion of subjects with HBsAg/Ab Seroconversion by Study Visit up to WEEK 48 (EES) | % Numbers of subjects with<br>HBsAg/Ab<br>Seroconversion/Numbers of<br>subjects with positive HBsAg and<br>Negative HBsAb at baseline | SAC [1] |
| 2.21. | FAS | Study specific | Proportion of subjects with HBeAg Loss by Study Visit up to WEEK 48/WEEK 96 (FAS) | %: Numbers of subjects with HBeAg loss/Numbers of subjects with positive HBeAg at baseline | SAC [1,2] |
| 2.22. | EES | Study specific | Proportion of subjects with HBeAg Loss by Study Visit up to WEEK 48 (EES) | %: Numbers of subjects with HBeAg loss/Numbers of subjects with positive HBeAg at baseline | SAC [1] |
| 2.23. | FAS | Study specific | Proportion of subjects with HBeAg/Ab Seroconversion by Study Visit up to WEEK 48/WEEK 96 (FAS) | % Numbers of subjects with HBeAg/Ab Seroconversion/Numbers of subjects with positive HBeAg and Negative HBeAb at baseline | SAC [1,2] |
| 2.24. | EES | Study specific | Proportion of subjects with HBeAg/Ab Seroconversion by Study Visit up to WEEK 48 (EES) | % Numbers of subjects with HBeAg/Ab Seroconversion/Numbers of subjects with positive HBeAg and Negative HBeAb at baseline | SAC [1] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Virolo | Virology | | | | |
| 2.25. | FAS | Study specific | Summary of HBcrAg by Study Visit up to WEEK 48/WEEK 96 (FAS) | Change from baseline is included. | SAC [1,2] |
| 2.26. | FAS | Study specific | Frequency of HBcrAg category by Study Visit up to WEEK 48/WEEK 96 (FAS) | HBcrAg category:<br><3.0 log10, 3.0<= - <4.0 log10,<br>4.0<= -<5.0 log10, 5.0<= - <6.0<br>log10, >=6.0 log10 Unit: KU/L | SAC [1,2] |
| 2.27. | FAS | Study specific | Proportion of subjects with HBV-DNA < 1.0 log10 IU/mL by Study Visit up to WEEK 48/WEEK 96 (FAS) | <1.0 log10 IU/mL, >=1.0 log10 IU/mL | SAC [1,2] |
| 2.28. | FAS | Study specific | Summary of HBV-DNA by Study Visit up to WEEK 48/WEEK 96 (FAS) | Change from baseline is included. | SAC [1,2] |
| 2.29. | FAS | Study specific | Summary of HBeAg by Study Visit up to WEEK 48 /WEEK 96 (FAS) | Change from baseline is included. | SAC [1,2] |
| 2.30. | FAS | Study specific | Summary of log10 HBeAg by Study Visit up to WEEK 48 /WEEK 96 (FAS) | Change from baseline is included. | SAC [1,2] |
| 2.31. | FAS | Study specific | Frequency of Virological Breakthrough (WEEK 0 – WEEK 48/WEEK 96) (FAS) | Change from baseline is included. | SAC [1,2] |
| 2.32. | FAS | Study specific | Summary of HBcrAg (Conventional unit) by Study Visit up to WEEK 48/WEEK 96 (FAS) | HBcrAg category:<br><3.0 log10, 3.0<= - <4.0 log10,<br>4.0<= -<5.0 log10, 5.0<= - <6.0<br>log10, >=6.0 log10 Unit: U/mL | SAC [1,2] |
| 2.33. | FAS | Study specific | Frequency of HBcrAg category (Conventional unit) by Study Visit up to WEEK 48/WEEK 96 (FAS) | | SAC [1,2] |
| ALT | | | | | |
| 2.34. | FAS | Study specific | Summary of ALT by Study Visit up to WEEK 48/WEEK 96 (FAS) | Change from baseline is included | SAC [1,2] |
| 2.35. | FAS | Study specific | Summary of ALT (Conventional unit) by Study Visit up to WEEK 48/WEEK 96 (FAS) | Change from baseline is included | SAC [1,2] |

| Effica | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subgre | Subgroup | | | | |
| 2.36. | FAS | Study specific | Summary of log10 HBsAg by Protocol defined liver cirrhosis (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.37. | FAS | Study specific | Summary of log10 HBsAg by Genotype (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.38. | FAS | Study specific | Summary of log10 HBsAg by HBsAg subgroup category (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.39. | FAS | Study specific | Summary of log10 HBsAg by AGE category (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.40. | FAS | Study specific | Summary of log10 HBsAg by Former Peg-INF (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.41. | FAS | Study specific | Summary of HBcrAg by Protocol defined liver cirrhosis (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.42. | FAS | Study specific | Summary of HBcrAg by Genotype (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.43. | FAS | Study specific | Summary of HBcrAg by HBsAg subgroup category (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.44. | FAS | Study specific | Summary of HBcrAg by AGE category (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.45. | FAS | Study specific | Summary of HBcrAg by Former Peg-INF (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.46. | FAS | Study specific | Summary of log10 HBeAg by Protocol defined liver cirrhosis (FAS, 48W/96W) | | SAC [1,2] |
| 2.47. | FAS | Study specific | Summary of log10 HBeAg by Genotype (FAS, 48W/96W) | | SAC [1,2] |
| 2.48. | FAS | Study specific | Summary of log10 HBeAg by HBsAg subgroup category (FAS, 48W/96W) | | SAC [1,2] |
| 2.49. | FAS | Study specific | Summary of log10 HBeAg by AGE category (FAS, 48W/96W) | | SAC [1,2] |

| Effica | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.50. | FAS | Study specific | Summary of log10 HBeAg by Former Peg-INF (FAS, 48W/96W) | | SAC [1,2] |
| 2.51. | FAS | Study specific | Summary of log10 HBsAg (Conventional unit) by Protocol defined liver cirrhosis (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.52. | FAS | Study specific | Summary of log10 HBsAg (Conventional unit) by Genotype (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.53. | FAS | Study specific | Summary of log10 HBsAg (Conventional unit) by HBsAg subgroup category (Conventional unit) (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.54. | FAS | Study specific | Summary of log10 HBsAg (Conventional unit) by AGE category (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.55. | FAS | Study specific | Summary of log10 HBsAg (Conventional unit) by Former Peg-INF (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.56. | FAS | Study specific | Summary of HBcrAg (Conventional unit) by Protocol defined liver cirrhosis (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.57. | FAS | Study specific | Summary of HBcrAg (Conventional unit) by Genotype (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.58. | FAS | Study specific | Summary of HBcrAg (Conventional unit) by HBsAg subgroup category (Conventional unit) (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.59. | FAS | Study specific | Summary of HBcrAg (Conventional unit) by AGE category (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.60. | FAS | Study specific | Summary of HBcrAg (Conventional unit) by Former Peg-INF (FAS, 48W/96W) | Change from baseline is included | SAC [1,2] |
| 2.61. | FAS | Study specific | Summary of log10 HBeAg by HBsAg subgroup category (Conventional unit) (FAS, 48W/96W) | | SAC [1,2] |

# 11.12.6. Efficacy Figures

| Effica | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| HBsA | HBsAg | | | | |
| 2.1. | FAS | Study specific | Log10 HBsAg by Study Visit up to WEEK 48/WEEK 96:<br>Mean (SD) Plots (FAS) | ± SD plots | SAC [1,2] |
| 2.2. | FAS | Study specific | Log10 HBsAg Change from Baseline by Study Visit up to WEEK 48/WEEK 96: Mean (SD) Plots (FAS) | ± SD plots | SAC [1,2] |
| 2.3. | FAS | Study specific | Log10 HBsAg (Conventional unit) by Study Visit up to WEEK 48/WEEK 96: Mean (SD) Plots (FAS) | ± SD plots | SAC [1,2] |
| 2.4. | FAS | Study specific | Log10 HBsAg (Conventional unit) Change from Baseline<br>by Study Visit up to WEEK 48/WEEK 96: Mean (SD)<br>Plots (FAS) | ± SD plots | SAC [1,2] |
| Virolo | gy | | | | |
| 2.5. | FAS | Study specific | HBcrAg by Study Visit up to WEEK 48/WEEK 96: Mean (SD) Plots (FAS) | ± SD plots | SAC [1,2] |
| 2.6. | FAS | Study specific | HBcrAg Change from Baseline by Study Visit up to WEEK 48/WEEK 96: Mean (SD) Plots (FAS) | ± SD plots | SAC [1,2] |
| 2.7. | FAS | Study specific | HBV-DNA by Study Visit up to WEEK 48/WEEK 96:<br>Mean (SD) Plots (FAS) | ± SD plots | SAC [1,2] |
| 2.8. | FAS | Study specific | HBV-DNA Change from Baseline by Study Visit up to WEEK 48/WEEK 96: Mean (SD) Plots (FAS) | ± SD plots | SAC [1,2] |
| 2.9. | FAS | Study specific | Log10 HBeAg Change from Baseline by Study Visit up to WEEK 48/WEEK 96: Mean (SD) Plots (FAS) | ± SD plots | SAC [1,2] |
| 2.10. | FAS | Study specific | HBcrAg (Conventional unit) by Study Visit up to WEEK 48/WEEK 96: Mean (SD) Plots (FAS) | ± SD plots | SAC [1,2] |
| 2.11. | FAS | Study specific | HBcrAg (Conventional unit) Change from Baseline by Study Visit up to WEEK 48/WEEK 96: Mean (SD) Plots (FAS) | ± SD plots | SAC [1,2] |

| Efficacy: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ALT | | | | | |
| 2.12. | FAS | Study specific | ALT by Study Visit up to WEEK 48/WEEK 96: Mean (SD) Plots (FAS) | ± SD plots | SAC [1,2] |
| 2.13. | FAS | Study specific | ALT Change from Baseline by Study Visit up to WEEK 48/WEEK 96: Mean (SD) Plots (FAS) | ± SD plots | SAC [1,2] |
| 2.14. | FAS | Study specific | ALT (Conventional unit) by Study Visit up to WEEK 48/WEEK 96: Mean (SD) Plots (FAS) | ± SD plots | SAC [1,2] |
| 2.15. | FAS | Study specific | ALT (Conventional unit) Change from Baseline by Study Visit up to WEEK 48/WEEK 96: Mean (SD) Plots (FAS) | ± SD plots | SAC [1,2] |

# 11.12.7. Safety Tables

| Safety | Safety: Tables | | | | | | |
|---|---|---|---|---|---|--|--|
| No. | Population | IDSL /<br>Example<br>Shell | Title | <b>Programming Notes</b> | Deliverable<br>[Priority] | | |
| Adver | se Events (AE | s) | | | · | | |
| 3.1. | Safety | AE1 | Summary of Adverse Events by System Organ Class and Preferred Term (WEEK 48/WEEK 96: on Treatment Period) | | SAC [1,2] | | |
| 3.2. | Safety | AE1 | Summary of Non-Serious Adverse Events by System Organ Class and Preferred Term, >=5% (WEEK 48/WEEK 96: on Treatment Period for FDAAA) | | SAC [1,2] | | |
| 3.3. | Safety | AE5A | Summary of Adverse Events by Maximum Intensity (WEEK 48/WEEK 96: on Treatment Period) | | SAC [1,2] | | |
| 3.4. | Safety | AE1 | Summary of Drug-Related Adverse Events by System Organ Class and Preferred Term (WEEK 48/WEEK 96: on Treatment Period) | | SAC [1,2] | | |
| 3.5. | Safety | AE5 | Summary of Drug-Related Adverse Events by Maximum Intensity (WEEK 48/WEEK 96: on Treatment Period) | | SAC [1,2] | | |
| 3.6. | Safety | AE1 | Summary of Adverse Events by 3 Months (WEEK 48 on Treatment Period) | | SAC [1] | | |
| 3.7. | Safety | AE1 | Summary of Adverse Events by 6 Months (WEEK 96 on Treatment Period) | | SAC [2] | | |
| Seriou | Serious and Other Significant Adverse Events | | | | | | |
| 3.8. | Safety | AE1 | Summary of Serious Adverse Events by System Organ<br>Class and Preferred Term (WEEK 48/WEEK 96: on<br>Treatment Period) | | SAC [1,2] | | |
| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.9. | Safety | AE1 | Summary of Fatal Serious Adverse Events by System Organ Class and Preferred Term (WEEK 48/WEEK 96: on Treatment Period) | | SAC [1,2] |
| 3.10. | Safety | AE1 | Summary of Adverse Events Leading to Permanent<br>Discontinuation of Study Drug by System Organ Class<br>and Preferred Term (WEEK 48/WEEK 96: on Treatment<br>Period) | | SAC [1,2] |
| AE of | Interest | | | | |
| 3.11. | Safety | AE1 | Summary of Renal AE as AE of Interest (WEEK 48/WEEK 96: on Treatment Period) | | SAC [1,2] |
| 3.12. | Safety | AE1 | Summary of Bone Events as AE of Interest (WEEK 48/WEEK 96: on Treatment Period) | | SAC [1,2] |
| 3.13. | Safety | AE1 | Summary of Liver AE as AE of Interest (WEEK 48/WEEK 96: on Treatment Period) | | SAC [1,2] |
| Labor | atory: Chemis | try | | | |
| 3.14. | Safety | LB1 | Summary of Chemistry Data | Change from baseline is included. Corrected calcium based on the serum albumin is included. Creatinine clearance is included. | SAC [1,2] |
| 3.15. | Safety | LB1 | Summary of Chemistry Results Relative to Normal Range | | SAC [1,2] |
| 3.16. | Safety | LB1 | Summary of Chemistry Data (ALT, ALP, Creatinine, Phosphorus, Glucose, Uric acid, eGFR) with conventional unit | Change from baseline is included. | SAC [1,2] |
| Labor | atory: Hemato | ology | | <u> </u> | |
| 3.17. | Safety | LB1 | Summary of Hematology Data | Change from baseline is included | SAC [1,2] |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.18. | Safety | LB1 | Summary of Hematology Results Relative to Normal Range | | SAC [1,2] |
| Labor | atory: Urinaly | vsis | | | • |
| 3.19. | Safety | UR3b | Summary of Urinalysis (Glucose, protein, urinary sediment,) Data | | SAC [1,2] |
| 3.20. | Safety | LB1 | Summary of Urinalysis (β2-microglobulin, β2-microglobulin-creatinine ratio, %TRP, creatinine, electrolyte (P)) | Change from baseline is included | SAC [1,2] |
| 3.21. | Safety | LB1 | Summary of Urinalysis ( $\beta$ 2-microglobulin, electrolyte (P), creatinine) with conventional unit | Change from baseline is included | SAC [1,2] |
| Labor | atory: Hepato | biliary (Liver) | | | • |
| 3.22. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | | SAC [1,2] |
| 3.23. | Safety | MH4 | Summary of Medical Conditions for Subjects with Liver<br>Stopping Events | | SAC [1,2] |
| 3.24. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | | SAC [1,2] |
| LDTA | GSI grade sc | ale | | | |
| 3.25. | Safety | Study specific | Summary of Treatment-Emergent Laboratory Abnormalities, LDTA GSI Grading Scale (WEEK 48/WEEK 96 on Treatment Period) | | SAC [1,2] |
| 3.26. | Safety | Study specific | Summary of LDTA GSI Grade 3/4 Treatment-Emergent Laboratory Abnormalities (WEEK 48/WEEK 96 on Treatment Period) | | SAC [1,2] |
| 3.27. | Safety | Study specific | Summary of Treatment-Emergent Marked Laboratory<br>Abnormalities, LDTA GSI Grading Scale (WEEK<br>48/WEEK 96 on Treatment Period) | See Section 11.6.4 safety, Gilead Science Institute (GSI) grading laboratory Data, Treatment-Emergent Marked Abnormalities | SAC [1,2] |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Hepati | c Flare | | | | |
| 3.28. | Safety | Study specific | Summary of On-Treatment Hepatic Flare (WEEK 48/WEEK 96 on Treatment Period) | | SAC [1,2] |
| 3.29. | Safety | Study specific | Summary of On-Treatment Laboratory Values Relevant to on-Treatment Hepatic Flare (WEEK 48/WEEK 96 on Treatment Period) | | SAC [1,2] |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Renal | Parameters | | | | |
| 3.30. | Safety | Study specific | Summary of Confirmed Changes in Renal Parameters (WEEK 48/WEEK 96 on treatment period) | | SAC [1,2] |
| GSI M | odified NIAII | D | | | |
| 3.31. | Safety | Study specific | Summary of Treatment-Emergent Laboratory Abnormalities, GSI Modified NIAID (WEEK 48/WEEK 96 on Treatment Period) | | SAC [1,2] |
| 3.32. | Safety | Study specific | Summary of GSI Modified NIAID Grade 3/4 Treatment-<br>Emergent Laboratory Abnormalities (WEEK 48/WEEK<br>96 on Treatment Period) | | SAC [1,2] |
| 3.33. | Safety | Study specific | Summary of Treatment-Emergent Marked Laboratory<br>Abnormalities, GSI Modified NIAID (WEEK 48/WEEK<br>96 on Treatment Period) | See Section 11.6.4 safety, Gilead Science Institute (GSI) grading laboratory Data, Treatment-Emergent Marked Abnormalities | SAC [1,2] |
| ECG | | | | | |
| 3.34. | Safety | EG1 | Summary of ECG Findings | | SAC [1,2] |
| 3.35. | Safety | EG2 | Summary of ECG Values | | SAC [1,2] |
| 3.36. | Safety | EG2 | Summary of Change from Baseline in ECG Values | | SAC [1,2] |
| Vital S | igns | | | | |
| 3.37. | Safety | VS1 | Summary of Vital Signs | | SAC [1,2] |
| 3.38. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | | SAC [1,2] |
| Others | | | | • | |
| 3.39. | Safety | VS1 | Summary of Percent Change from Baseline in Bone<br>Density (DEXA method: %) by position | | SAC [1,2] |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.40. | Safety | VS1 | Summary of Bone Density (DEXA method: absolute) by position | Change from baseline is included. | SAC [1,2] |

# 11.12.8. Safety Figures

| Safety | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | <b>Programming Notes</b> | Deliverable<br>[Priority] |
| Labor | atory: Chemis | stry | | | |
| 3.1. | Safety | Study specific | Creatinine by Study Visit: Mean (SD) Plots | ± SD plots | SAC [1,2] |
| 3.2. | Safety | Study specific | Creatinine Change from Baseline by Study Visit: Mean (SD) Plots | ± SD plots | SAC [1,2] |
| 3.3. | Safety | Study specific | eGFR by Study Visit: Mean (SD) Plots | ± SD plots | SAC [1,2] |
| 3.4. | Safety | Study specific | eGFR Change from Baseline by Study Visit: Mean (SD)<br>Plots | ± SD plots | SAC [1,2] |
| 3.5. | Safety | Study specific | Creatinine (Conventional unit) by Study Visit: Mean (SD) Plots | ± SD plots | SAC [1,2] |
| 3.6. | Safety | Study specific | Creatinine (Conventional unit) Change from Baseline with conventional unit by Study Visit: Mean (SD) Plots | ± SD plots | SAC [1,2] |
| 3.7. | Safety | Study specific | eGFR (Conventional unit) by Study Visit: Mean (SD)<br>Plots | ± SD plots | SAC [1,2] |
| 3.8. | Safety | Study specific | eGFR (Conventional unit) Change from Baseline by<br>Study Visit: Mean (SD) Plots | ± SD plots | SAC [1,2] |
| Labor | atory: Other | | | | |
| 3.9. | Safety | Study specific | Bone Density (DEXA method, absolute) by position:<br>Mean (SD) Plots for change from baseline | DEXA method ± SD plots | SAC [1,2] |
| 3.10. | Safety | Study specific | Bone Density (DEXA method, %) by position: Mean (SD) Plots for %change from baseline | DEXA method ± SD plots | SAC [1,2] |

#### 11.12.9. Exploratory Statistical Analysis Tables

| Explo | Exploratory Statistical Analysis Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| HBsA | g Responder/N | on-Responder | | | • |
| 4.1. | FAS | Study specific | Frequency of HBsAg Responder/Non-responder with ALT category (<60 IU/L, >=60IU/L) at WEEK 48 | | SAC [1] |
| 4.2. | FAS | Study specific | Frequency of HBsAg Responder/Non-responder with ALT category (Conventional unit) (<60 U/L, >=60U/L) at WEEK 48 | | SAC [1] |
| HBsA | g Responder/N | on-Responder: | HBsAg | | |
| 4.3. | FAS | Study specific | Summary of log10 HBsAg during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder (FAS) | Change from baseline is included | SAC [1,2] |
| 4.4. | FAS | Study specific | Summary of log10 HBsAg (Conventional unit) during<br>Study Visit up to WEEK 48/WEEK 96 by HBsAg<br>Responder / Non-responder (FAS) | Change from baseline is included | SAC [1,2] |
| HBsA | g Responder/N | on-Responder: | Other Efficacy | | • |
| 4.5. | FAS | Study specific | Summary of HBcrAg during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder (FAS) | Change from baseline is included | SAC [1,2] |
| 4.6. | FAS | Study specific | Summary of HBV-DNA during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder (FAS) | Change from baseline is included | SAC [1,2] |
| 4.7. | FAS | Study specific | Summary of ALT during Study Visit up to WEEK<br>48/WEEK 96 by HBsAg Responder / Non-responder<br>(FAS) | Change from baseline is included | SAC [1,2] |
| 4.8. | FAS | Study specific | Summary of ALT category (<60 IU/L, >=60 IU/L) during<br>Study Visit up to WEEK 48/WEEK 96 by HBsAg<br>Responder / Non-responder (FAS) | | SAC [1,2] |

| Explo | Exploratory Statistical Analysis Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.9. | FAS | Study specific | Summary of log10 HBeAg during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder (FAS) | Change from baseline is included | SAC [1,2] |
| 4.10. | FAS | Study specific | Summary of HBcrAg (Conventional unit) during Study<br>Visit up to WEEK 48/WEEK 96 by HBsAg Responder /<br>Non-responder (FAS) | Change from baseline is included | SAC [1,2] |
| 4.11. | FAS | Study specific | Summary of ALT (Conventional unit) during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder (FAS) | Change from baseline is included | SAC [1,2] |
| 4.12. | FAS | Study specific | Summary of ALT category (Conventional unit) (<60 U/L, >=60 U/L) during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder (FAS) | | SAC [1,2] |
| ALT ( | Category (<60 | IU/L, >=60 IU/L | ): HBsAg | | |
| 4.13. | FAS | Study specific | Summary of log10 HBsAg during Study Visit up to WEEK 48/WEEK 96 by ALT Category (<60IU/L, >=60IU/L) (FAS) | Change from baseline is included | SAC [1,2] |
| 4.14. | FAS | Study specific | Summary of log10 HBsAg (Conventional unit) during<br>Study Visit up to WEEK 48/WEEK 96 by ALT Category<br>(Conventional unit) (<60U/L, >=60U/L) (FAS) | Change from baseline is included | SAC [1,2] |
| ALT ( | Category (<60 | IU/L, >=60 IU/L | ): Other Efficacy | | |
| 4.15. | FAS | Study specific | Summary of HBcrAg during Study Visit up to WEEK 48/WEEK 96 by ALT Category (<60 IU/L, >=60I U/L) (FAS) | Change from baseline is included | SAC [1,2] |
| 4.16. | FAS | Study specific | Summary HBV-DNA during Study Visit up to WEEK 48/WEEK 96 by ALT Category (<60 IU/L, >=60 IU/L) (FAS) | Change from baseline is included | SAC [1,2] |
| 4.17. | FAS | Study specific | Summary of ALT during Study Visit up to WEEK 48/WEEK 96 by ALT Category (<60 IU/L, >=60 IU/L) (FAS) | Change from baseline is included | SAC [1,2] |

| Explo | Exploratory Statistical Analysis Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.18. | FAS | Study specific | Summary of log10 HBeAg during Study Visit up to WEEK 48/WEEK 96 by ALT Category (<60 IU/L, >=60 IU/L) (FAS) | Change from baseline is included | SAC [1,2] |
| ALT ( | Category (<60 | U/L, >=60 U/L): | Other Efficacy | | |
| 4.19. | FAS | Study specific | Summary of HBcrAg (Conventional unit) during Study Visit up to WEEK 48/WEEK 96 by ALT Category (Conventional unit) (<60 U/L, >=60 U/L) (FAS) | Change from baseline is included | SAC [1,2] |
| 4.20. | FAS | Study specific | Summary HBV-DNA during Study Visit up to WEEK 48/WEEK 96 by ALT Category (Conventional unit) (<60 U/L, >=60 U/L) (FAS) | Change from baseline is included | SAC [1,2] |
| 4.21. | FAS | Study specific | Summary of ALT (Conventional unit) during Study Visit up to WEEK 48/WEEK 96 by ALT Category (Conventional unit) (<60 U/L, >=60 U/L) (FAS) | Change from baseline is included | SAC [1,2] |
| 4.22. | FAS | Study specific | Summary of log10 HBeAg during Study Visit up to WEEK 48/WEEK 96 by ALT Category (Conventional unit) (<60 U/L, >=60 U/L) (FAS) | Change from baseline is included | SAC [1,2] |
| Backg | round of HBsA | Ag Responder/ N | on-Responder: Demographic and Baseline Characteristic | es | |
| 4.23. | FAS | DM1 | Summary of Demographic Characteristics by HBsAg<br>Responder / Non-responder (FAS) | | SAC [1] |
| 4.24. | FAS | Study specific | Summary of Other Baseline Characteristics by HBsAg<br>Responder / Non-responder (FAS) | | SAC [1] |
| Backg | round of HBsA | Ag Responder/ N | on-Responder: Medical Conditions and Concomitant Me | dications | |
| 4.25. | FAS | MH4 | Summary of Prior Medical Conditions by HBsAg<br>Responder / Non-responder (FAS) | | SAC [1] |
| 4.26. | FAS | CM1 | Summary of Concomitant Medications by HBsAg<br>Responder / Non-responder (FAS) | | SAC [1] |
| Backg | round of HBsA | Ag Responder/ N | on-Responder: Exposure and Treatment Compliance | | • |
| 4.27. | FAS | Study specific | Summary of Treatment Compliance by HBsAg<br>Responder / Non-responder (FAS) | | SAC [1] |

| Explo | Exploratory Statistical Analysis Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | <b>Programming Notes</b> | Deliverable<br>[Priority] |
| 4.28. | FAS | EX1 | Duration of Exposure to Study Drug by HBsAg<br>Responder / Non-responder(FAS) | | SAC [1] |
| Safety | Subgroup An | alysis | | | |
| 4.29. | Safety | Study specific | Summary of eGFR by Subgroup (SP) | AGE category (<40, 40-49, 50-59, 60-), eGFR baseline category (<1, 1<= - <1.5, >=1.5), Weight baseline category (<50 kg, >=50 kg), Sex (male, female) | SAC [1,2] |
| 4.30. | Safety | Study specific | Summary of Beta2-microglobulin-creatinine ratio by Subgroup (SP) | AGE category (<40, 40-49, 50-59, 60-), eGFR baseline category (<1, 1<= - <1.5, >=1.5), Weight baseline category (<50 kg, >=50 kg), Sex (male, female) | SAC [1,2] |
| 4.31. | Safety | Study specific | Summary of %TRP by Subgroup (SP) | AGE category (<40, 40-49, 50-59, 60-), eGFR baseline category (<1, <=1-<1.5, >=1.5), Weight baseline category (<50 kg, >=50 kg), Sex (male, female) | SAC [1,2] |
| 4.32. | Safety | Study specific | Summary of Serum Creatine by Subgroup (SP) | AGE category (<40, 40-49, 50-59, 60-), eGFR baseline category (<1, 1<= - <1.5, >=1.5), Weight baseline category (<50 kg, >=50 kg), Sex (male, female) | SAC [1,2] |
| 4.33. | Safety | Study specific | Summary of Serum Phosphorus by Subgroup (SP) | AGE category (<40, 40-49, 50-59, 60-), eGFR baseline category (<1, 1<= - <1.5, >=1.5), Weight baseline category (<50 kg, >=50 kg), Sex (male, female) | SAC [1,2] |

| Explo | Exploratory Statistical Analysis Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.34. | Safety | Study specific | Summary of Bone density(absolute) by Subgroup (SP) | Change from baseline is included.<br>AGE category (<40, 40-49, 50-59, 60-), eGFR baseline category (<1, 1<= - <1.5, >=1.5), Weight baseline category (<50 kg, >=50 kg), Sex (male, female) | SAC [1,2] |
| 4.35. | Safety | Study specific | Summary of Bone density (%change from baseline) by Subgroup (SP) | AGE category (<40, 40-49, 50-59, 60-), eGFR baseline category (<1, 1<= - <1.5, >=1.5), Weight baseline category (<50 kg, >=50 kg), Sex (male, female) | SAC [1,2] |
| 4.36. | Safety | Study specific | Summary of eGFR (Conventional unit) by Subgroup (SP) | AGE category (<40, 40-49, 50-59, 60-), eGFR baseline category (<60, 60<= - <90, >=90), Weight baseline category (<50 kg, >=50 kg), Sex (male, female) | SAC [1,2] |
| 4.37. | Safety | Study specific | Summary of Beta2-microglobulin-creatinine ratio by Subgroup (SP) | AGE category (<40, 40-49, 50-59, 60-), eGFR baseline category (<60, 60<= - <90, >=90), Weight baseline category (<50 kg, >=50 kg), Sex (male, female) | SAC [1,2] |
| 4.38. | Safety | Study specific | Summary of %TRP by Subgroup (SP) | AGE category (<40, 40-49, 50-59, 60-), eGFR baseline category (<60, 60 <= - <90 >=90), Weight baseline category (<50 kg, >=50 kg), Sex (male, female) | SAC [1,2] |
| 4.39. | Safety | Study specific | Summary of Serum Creatine (Conventional unit) by Subgroup (SP) | AGE category (<40, 40-49, 50-59, 60-), eGFR baseline category (<60, 60<= - <90, >=90), Weight baseline category (<50 kg, >=50 kg), Sex (male, female) | SAC [1,2] |

| Explo | Exploratory Statistical Analysis Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.40. | Safety | Study specific | Summary of Serum Phosphorous (Conventional unit) by Subgroup (SP) | AGE category (<40, 40-49, 50-59, 60-), eGFR baseline category (<60, 60<= - <90, >=90), Weight baseline category (<50 kg, >=50 kg), Sex (male, female) | SAC [1,2] |
| 4.41. | Safety | Study specific | Summary of Bone density(absolute) by Subgroup (SP) | Change from baseline is included. AGE category (<40, 40-49, 50-59, 60-), eGFR baseline category (<60, 60<= - <90, >=90), Weight baseline category (<50 kg, >=50 kg), Sex (male, female) | SAC [1,2] |
| 4.42. | Safety | Study specific | Summary of Bone density (%change from baseline) by Subgroup (SP) | AGE category (<40, 40-49, 50-59, 60-), eGFR baseline category (<60, 60<= - <90, >=90), Weight baseline category (<50 kg, >=50 kg), Sex (male, female) | SAC [1,2] |

## 11.12.10. Exploratory Statistical Analysis Figures

| Explor | Exploratory Statistical Analysis Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| HBsAg | g Responder/No | n-Responder: 1 | HBsAg | | • |
| 4.1. | FAS | Study specific | Log10 HBsAg during Study Visit up to WEEK<br>48/WEEK 96 by HBsAg Responder / Non-responder:<br>Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.2. | FAS | Study specific | Log10 HBsAg Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder: Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.3. | FAS | Study specific | Log10 HBsAg Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder: Individual Plots (FAS) | | SAC [1,2] |
| HBsAg | g Responder/No | n-Responder: 1 | HBsAg (Conventional unit) | | • |
| 4.4. | FAS | Study specific | Log10 HBsAg (Conventional unit) during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder: Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.5. | FAS | Study specific | Log10 HBsAg (Conventional unit) Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder: Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.6. | FAS | Study specific | Log10 HBsAg (Conventional unit) Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder: Individual Plots (FAS) | | SAC [1,2] |
| HBsAg | g Responder/No | n-Responder: ( | | | _ |
| 4.7. | FAS | Study specific | HBcrAg during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder: Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.8. | FAS | Study specific | HBcrAg Change from Baseline during Study Visit up to WEEK 48 /WEEK 96 by HBsAg Responder / Non-responder: Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |

| Explor | Exploratory Statistical Analysis Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.9. | FAS | Study specific | HBV-DNA during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder: Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.10. | FAS | Study specific | HBV-DNA Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder: Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.11. | FAS | Study specific | ALT during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder, Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.12. | FAS | Study specific | ALT Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder: Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.13. | FAS | Study specific | Log10 HBeAg during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder; Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.14. | FAS | Study specific | Log10 HBeAg Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder: Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| HBsAg | Responder/No | n-Responder: | Other Efficacy (Conventional unit) | | |
| 4.15. | FAS | Study specific | HBcrAg (Conventional unit) during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder: Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.16. | FAS | Study specific | HBcrAg (Conventional unit) Change from Baseline during Study Visit up to WEEK 48 /WEEK 96 by HBsAg Responder / Non-responder: Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.17. | FAS | Study specific | ALT (Conventional unit) during Study Visit up to WEEK 48/WEEK 96 by HBsAg Responder / Non-responder, Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |

| Explor | Exploratory Statistical Analysis Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.18. | FAS | Study specific | ALT (Conventional unit) Change from Baseline during<br>Study Visit up to WEEK 48/WEEK 96 by HBsAg<br>Responder / Non-responder: Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| ALT C | ategory (<60 II | U/L, >=60 IU/L) | | | |
| 4.19. | FAS | Study specific | Log10 HBsAg during Study Visit up to WEEK<br>48/WEEK 96 by ALT Category (<60 IU/L, >=60 IU/L):<br>Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.20. | FAS | Study specific | Log10 HBsAg Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by ALT Category (<60 IU/L, >=60 IU/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| ALT C | ategory (<60 U | /L, >=60 U/L): | HBsAg (Conventional unit) | | |
| 4.21. | FAS | Study specific | Log10 HBsAg (Conventional unit) during Study Visit up to WEEK 48/WEEK 96 by ALT Category (Conventional unit) (<60 U/L, >=60 U/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.22. | FAS | Study specific | Log10 HBsAg (Conventional unit) Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by ALT Category (Conventional unit) (<60 U/L, >=60 U/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| ALT C | ategory (<60 II | U/L, >=60 IU/L) | ): Other Efficacy | | |
| 4.23. | FAS | Study specific | HBcrAg during Study Visit up to WEEK 48/WEEK 96 by ALT Category (<60 IU/L, >=60 IU/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.24. | FAS | Study specific | HBcrAg Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by ALT Category (<60 IU/L, >=60 IU/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.25. | FAS | Study specific | HBV-DNA during Study Visit up to WEEK 48/WEEK 96 by ALT Category (<60 IU/L, >=60 IU/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |

| Explor | Exploratory Statistical Analysis Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.26. | FAS | Study specific | HBV-DNA Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by ALT Category (<60 IU/L, >=60 IU/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.27. | FAS | Study specific | ALT during Study Visit up to WEEK 48/WEEK 96 by ALT Category (<60 IU/L, >=60 IU/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.28. | FAS | Study specific | ALT Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by ALT Category (<60 IU/L, >=60 IU/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.29. | FAS | Study specific | Log10 HBeAg during Study Visit up to WEEK<br>48/WEEK 96 by ALT Category (<60 IU/L, >=60 IU/L):<br>Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.30. | FAS | Study specific | Log10 HBeAg Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by ALT Category (<60 IU/L, >=60 IU/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| ALT C | ategory (<60 U | I/L, >=60 U/L): | Other Efficacy (Conventional unit) | | |
| 4.31. | FAS | Study specific | HBcrAg (Conventional unit) during Study Visit up to WEEK 48/WEEK 96 by ALT Category (Conventional unit) (<60 U/L, >=60 U/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.32. | FAS | Study specific | HBcrAg (Conventional unit) Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by ALT Category (Conventional unit) (<60 U/L, >=60 U/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.33. | FAS | Study specific | HBV-DNA during Study Visit up to WEEK 48/WEEK 96 by ALT Category (Conventional unit) (<60 U/L, >=60 U/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.34. | FAS | Study specific | HBV-DNA Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by ALT Category (Conventional unit) (<60 U/L, >=60 U/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |

| Explor | Exploratory Statistical Analysis Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.35. | FAS | Study specific | ALT (Conventional unit) during Study Visit up to WEEK 48/WEEK 96 by ALT Category (Conventional unit) (<60 U/L, >=60 U/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.36. | FAS | Study specific | ALT (Conventional unit) Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by ALT Category (Conventional unit) (<60 U/L, >=60 U/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.37. | FAS | Study specific | Log10 HBeAg during Study Visit up to WEEK 48/WEEK 96 by ALT Category (Conventional unit) (<60 U/L, >=60 U/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| 4.38. | FAS | Study<br>specific | Log10 HBeAg Change from Baseline during Study Visit up to WEEK 48/WEEK 96 by ALT Category (Conventional unit) (<60 U/L, >=60 U/L): Mean (SD) Plots (FAS) | ± SD plot | SAC [1,2] |
| Correl | ation of virus p | arameters | | | |
| 4.39. | FAS | Study specific | Log10 HBsAg Change from Baseline vs ALT Change from Baseline at WEEK24/WEEK 48/WEEK 96 (FAS) | X axis:Log10 HBsAg Change from Baseline | SAC [1,2] |
| 4.40. | FAS | Study<br>specific | Log10 HBsAg Change from Baseline vs HBcrAg<br>Baseline at WEEK24/WEEK 48/WEEK 96 (FAS) | X axis:Log10 HBsAg Change from Baseline | SAC [1,2] |
| 4.41. | FAS | Study<br>specific | Log10 HBsAg Change from Baseline vs HBcrAg Change from Baseline at WEEK24/WEEK 48/WEEK 96 (FAS) | X axis:Log10 HBsAg Change from Baseline | SAC [1,2] |
| 4.42. | FAS | Study specific | Log10 HBsAg Change from Baseline vs log10 HBeAg<br>Baseline at WEEK24/WEEK 48/WEEK 96 (FAS) | X axis:Log10 HBsAg Change from Baseline | SAC [1,2] |
| 4.43. | FAS | Study specific | Log10 HBsAg Change from Baseline vs log10 HBeAg<br>Change from Baseline at WEEK24/WEEK 48/WEEK 96<br>(FAS) | X axis:Log10 HBsAg Change from Baseline | SAC [1,2] |

| Explor | Exploratory Statistical Analysis Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | <b>Programming Notes</b> | Deliverable<br>[Priority] |
| Correla | ation of virus p | arameters (Con | ventional unit) | | |
| 4.44. | FAS | Study specific | Log10 HBsAg (Conventional unit) Change from Baseline vs ALT (Conventional unit) Change from Baseline at WEEK24/WEEK 48/WEEK 96 (FAS) | X axis:Log10 HBsAg<br>(Conventional unit) Change from<br>Baseline | SAC [1,2] |
| 4.45. | FAS | Study specific | Log10 HBsAg (Conventional unit) Change from Baseline vs HBcrAg (Conventional unit) Baseline at WEEK24/WEEK 48/WEEK 96 (FAS) | X axis:Log10 HBsAg<br>(Conventional unit) Change from<br>Baseline | SAC [1,2] |
| 4.46. | FAS | Study specific | Log10 HBsAg (Conventional unit) Change from Baseline vs HBcrAg (Conventional unit) Change from Baseline at WEEK24/WEEK 48/WEEK 96 (FAS) | X axis:Log10 HBsAg<br>(Conventional unit) Change from<br>Baseline | SAC [1,2] |
| 4.47. | FAS | Study specific | Log10 HBsAg (Conventional unit) Change from Baseline vs log10 HBeAg Baseline at WEEK24/WEEK 48/WEEK 96 (FAS) | X axis:Log10 HBsAg<br>(Conventional unit) Change from<br>Baseline | SAC [1,2] |
| 4.48. | FAS | Study specific | Log10 HBsAg (Conventional unit) Change from Baseline vs log10 HBeAg Change from Baseline at WEEK24/WEEK 48/WEEK 96 (FAS) | X axis:Log10 HBsAg<br>(Conventional unit) Change from<br>Baseline | SAC [1,2] |

#### **11.12.11.** ICH Listings

| ICH: | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject Disposition | | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | | SAC [1,2] |
| 2. | Safety | ES2 | Listing of Reasons for Study Withdrawal | | SAC [1,2] |
| 3. | Safety | SD2 | Listing of Reasons for Study Treatment Discontinuation | | SAC [1,2] |
| Protoc | Protocol Deviations | | | | |
| 4. | Safety | DV2 | Listing of Important Protocol Deviations | | SAC [1,2] |
| 5. | Screened | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | | SAC [1,2] |
| Popula | ations Analysed | | | | |
| 6. | Safety | SP3 | Listing of Subjects Excluded from EES Population (48W) | | SAC [1] |
| Demog | graphic and Base | eline Character | istics | | |
| 7. | Safety | DM2 | Listing of Demographic Characteristic | "Age at Screening" is added. | SAC [1,2] |
| 8. | Screening<br>Failure | DM2 | Listing of Demographic Characteristics for Screening Failure Subjects | | SAC [1] |
| 9. | Safety | DM9 | Listing of Race | | SAC [1,2] |
| 10. | Screening<br>Failure | DM9 | Listing of Race for Screening Failure Subjects | Treatment is not needed to display. | SAC [1] |
| 11. | Safety | Study specific | Listing of Other Baseline Characteristics | | SAC [1,2] |

| ICH: | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Medic | Medical Conditions and Concomitant Medications | | | | |
| 12. | Safety | MH2 | Listing of Medical Conditions (48W/96W) | | SAC [1,2] |
| 13. | Safety | CM3 | Listing of Prior Hepatitis Medications | | SAC [1] |
| 14. | Safety | CM3 | Listing of Concomitant Medications (48W/96W) | | SAC [1,2] |
| Expos | ure and Treatm | ent Compliance | | | |
| 15. | Safety | Study<br>specific | Listing of Treatment Compliance (48W/96W) | | SAC [1,2] |
| 16. | Safety | EX3 | Listing of Exposure Data (48W/96W) | | SAC [1,2] |
| Effica | cy: HBsAg | | | | |
| 17. | FAS | Study<br>specific | Listing of Efficacy Data (HBsAg Responder) | Log10 HBsAg Change from Baseline is included. | SAC [1,2] |
| 18. | FAS | Study<br>specific | Listing of Efficacy Data (log10 HBsAg) | Change from Baseline is included. | SAC [1,2] |
| 19. | FAS | Study<br>specific | Listing of Efficacy Data (HBsAg) | Change from Baseline is included. | SAC [1,2] |
| 20. | FAS | Study<br>specific | Listing of Efficacy Data (log10 HBsAg: Conventional unit) | Change from Baseline is included. | SAC [1,2] |
| 21. | FAS | Study<br>specific | Listing of Efficacy Data (HBsAg: Conventional unit) | Change from Baseline is included. | SAC [1,2] |
| Effica | cy: Seroconversi | on | | | |
| 22. | FAS | Study<br>specific | Listing of Efficacy Data (HBsAg) | Include POS/NEG data. | SAC [1,2] |

| ICH: | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 23. | FAS | Study<br>specific | Listing of Efficacy Data (HBsAb) | | SAC [1,2] |
| 24. | FAS | Study specific | Listing of Efficacy Data (HBeAg) | Include POS/NEG data log 10 HBeAg is included | SAC [1,2] |
| 25. | FAS | Study specific | Listing of Efficacy Data (HBeAb) | | SAC [1,2] |
| Effica | cy: Virology | | | | |
| 26. | FAS | Study specific | Listing of Efficacy Data (HBcrAg) | Change from Baseline is included. | SAC [1,2] |
| 27. | FAS | Study specific | Listing of Efficacy Data (HBV-DNA) | log10 HBV-DNA data, log10<br>HBV-DNA Change from Baseline<br>is included. | SAC [1,2] |
| 28. | FAS | Study<br>Specifics | Listing of Efficacy Data (Virologic Breakthrough) | Virological breakthrough has been observed (a case where the serum HBV-DNA level has increased from the nadir by at least 1 log IU/mL, or HBV DNA level has increased to ≥2 log IU/mL (100 IU/mL) in a case with nadir <10 IU/mL) from Day1 to WEEK48/WEEK96. | SAC [1,2] |
| 29. | FAS | Study<br>specific | Listing of Efficacy Data (HBcrAg: Conventional unit) | Change from Baseline is included. | SAC [1,2] |
| Effica | Efficacy: ALT | | | | |
| 30. | FAS | Study specific | Listing of Efficacy Data (ALT) | Change from Baseline is included. | SAC [1,2] |

| ICH: | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 31. | FAS | Study specific | Listing of Efficacy Data (ALT: Conventional unit) | Change from Baseline is included. | SAC [1,2] |
| Adver | se Events | | | | |
| 32. | Safety | AE8 | Listing of All Adverse Events | | SAC [1,2] |
| 33. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse<br>Events | | SAC [1,2] |
| 34. | Safety | AE2 | Listing of Relationship Between Adverse Event System<br>Organ Classes, Preferred Terms, and Verbatim Text | | SAC [1,2] |
| Seriou | s Adverse Event | S | | | |
| 35. | Safety | AE8 | Listing of Serious Adverse Events | | SAC [1,2] |
| 36. | Safety | AE8 | Listing of Fatal Serious Adverse Events | | SAC [1,2] |
| Other | significant Adve | erse Events | | | |
| 37. | Safety | AE8 | Listing of Other Significant Adverse Events Leading to Withdrawal from Study | | SAC [1,2] |
| AE of | interest | | | | |
| 38. | Safety | AE8 | Listing of Renal AE as AE of Interest | | SAC [1,2] |
| 39. | Safety | AE8 | Listing of Bone Events as AE of Interest | | SAC [1,2] |
| 40. | Safety | AE8 | Listing of Liver AE as AE of Interest | | SAC [1,2] |
| Clinic | al Laboratory: C | Chemistry | | | |
| 41. | Safety | LB5 | Listing of All Chemistry Data | Change from Baseline is included. Corrected calcium based on the serum albumin is included. | SAC [1,2] |

| ICH: | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 42. | Safety | LB5 | Listing of Chemistry Data (ALT, ALP, Creatinine, Phosphorus, Glucose, Uric acid, eGFR) with conventional unit | Change from baseline is included. | SAC [1,2] |
| Clinic | al Laboratory: I | Hematology | | | |
| 43. | Safety | LB5 | Listing of All Hematology Data | Change from Baseline is included. | SAC [1,2] |
| Clinic | al Laboratory: <b>U</b> | Jrinalysis | | | |
| 44. | Safety | LB14 | Listing of Urinalysis (Glucose, protein, urinary sediment,) Data | | SAC [1,2] |
| 45. | Safety | UR2A | Listing of Urinalysis (β2-microglobulin, β2-microglobulin-creatinine ratio, %TRP, creatinine, electrolyte (P)) | Change from Baseline is included. | SAC [1,2] |
| 46. | Safety | URA2 | Listing of Urinalysis (β2-microglobulin, electrolyte (P), creatinine) with conventional unit | Change from baseline is included | SAC [1,2] |
| Hepat | obiliary (Liver) | - | | , | |
| 47. | Safety | Liver5 | Listing of Liver Monitoring/Stopping Event Reporting | IDSL | SAC [1,2] |
| 48. | Safety | MH2 | Listing of Medical Conditions for Participants with Liver<br>Stopping Events | IDSL | SAC [1,2] |
| 49. | Safety | Liver13 | Listing of Hepatobiliary Laboratory Abnormalities | IDSL | SAC [1,2] |
| LDTA | GSI grade scale | e | | | |
| 50. | Safety | LB5 | Listing of Treatment-Emergent Laboratory Abnormalities (LDTA GSI grade) | Include Marked Laboratory<br>Abnormalities | SAC [1,2] |
| 51. | Safety | LB5 | Listing of LDTA GSI Grade 3/4 Treatment-Emergent Laboratory Abnormalities | | SAC [1,2] |
| 52. | Safety | LB5 | Listing of All Hematology Data with LDTA GSI Grade | | SAC [1,2] |

| ICH: | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 53. | Safety | LB5 | Listing of All Chemistry Data with LDTA GSI Grade | | SAC [1,2] |
| Hepati | c Flare | | | | |
| 54. | Safety | Study<br>specific | Listing of on-Treatment Hepatic Flare | | SAC [1,2] |
| 55. | Safety | Study specific | Listing of On-Treatment Laboratory Values Relevant to On-Treatment Hepatic Flare | | SAC [1,2] |
| Renal | Parameters | | | | · |
| 56. | Safety | LB5 | Listing of Subjects with Cond Serum Creatinine Increase of 0.5 mg/dL Above Baseline (or Last Value on Drug) | | SAC [1,2] |
| 57. | Safety | LB5 | Listing of Subjects with Confirmed Serum Phosphorus <= 2 mg/dL (or Last Value on Drug) | | SAC [1,2] |
| 58. | Safety | LB5 | Listing of Subjects with Confirmed Creatinine Clearance < 50 mL/min (or Last Value on Drug) | | SAC [1,2] |
| GSI M | odified NIAID | | | | |
| 59. | Safety | Study specific | Listing of Treatment-Emergent Laboratory Abnormalities (GSI Modified NIAID) | Include Marked Laboratory<br>Abnormalities | SAC [1,2] |
| 60. | Safety | Study<br>specific | Listing of Grade 3/4 Treatment-Emergent Laboratory<br>Abnormalities (GSI Modified NIAID) | | SAC [1,2] |
| 61. | Safety | LB5 | Listing of All Hematology Data with GSI Modified NIAID | | SAC [1,2] |
| 62. | Safety | LB5 | Listing of All Chemistry Data with GSI Modified NIAID | | SAC [1,2] |
| ECG | | | | | |
| 63. | Safety | EG3 | Listing of All ECG Values | | SAC [1,2] |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 64. | Safety | EG3 | Listing of Change from Baseline in ECG Values | Listing will be divided as 64.1 and 64.2 | SAC [1,2] |
| 65. | Safety | EG5 | Listing of ECG Findings | Listing will be divided as 65.1 and 65.2 | SAC [1,2] |
| Vital Signs | | | | | |
| 66. | Safety | VS4 | Listing of All Vital Signs | | SAC [1,2] |
| 67. | Safety | VS4 | Listing of Change from Baseline in Vital Signs | | SAC [1,2] |
| Others | | | | | |
| 68. | Safety | Study specific | Listing of All Bone density for %change from Baseline | include all method and position. | SAC [1,2] |
| 69. | Safety | Study<br>specific | Listing of All Bone density (Absolute) | include all method and position. | SAC [1,2] |
| Explanatory Statistical Analysis | | | | | |
| 70. | Safety | Study<br>specific | Listing of subject numbers for individual HBsAg<br>Responder/Non-Responder Category at WEEK<br>48/WEEK 96 | | SAC [1,2] |
| 71. | Safety | Study<br>specific | Listing of subject numbers for individual ALT Category (<60 IU/L, >=60 IU/L) at WEEK 48/WEEK 96 | | SAC [1,2] |
| 72. | Safety | Study<br>specific | Listing of subject numbers for individual ALT Category (Conventional unit) (<60 U/L, >=60 U/L) at WEEK 48/WEEK 96 | | SAC [1,2] |

## 11.13. Appendix 13: Example Mock Shells for Data Displays

Mock-up displays will be provided separately.